# STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Placebo-Controlled, Dose Assessment Phase 2 Study to Evaluate the Safety and Efficacy of CCX168 in Subjects with Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis

Protocol Number: CL003 168

Investigational Product: Complement 5a Receptor Antagonist CCX168

Sponsor:

ChemoCentryx, Inc.

PPD

Version Number 1.0

Date: April 1, 2016

### CONFIDENTIAL

The information contained herein is the property of the Sponsor and may not be reproduced, published, or disclosed to others without the written authorization from the Sponsor.

# SIGNATURE PAGE

Protocol Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Assessment Phase 2 Study to Evaluate the Safety and Efficacy of CCX168 in Subjects with Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis

| Signature | Date |
|---------------------------------------------|-------------|
| PPD | 1-A4R-2016 |
| Chief Medical Officer<br>ChemoCentryx, Inc. | |
| PPD | 1- Apr-2016 |
| Biostatistician<br>PPD | |
| PPD | 04 apr 2016 |
| Medical Monitor | |

# REVISION HISTORY

| Version | Date | Description of Changes |
|---------|---------------|------------------------|
| 1.0 | April 1, 2016 | Original SAP |

# TABLE OF CONTENTS

| 1 | Intro | oduction | . 5 |
|---|-------|-----------------------------------------------------|-----|
| 2 | Tria | d Objectives | . 5 |
| 3 | Stat | ristical Methodology | . 6 |
| | 3.1 | Analysis Populations | . 6 |
| | 3.2 | Analysis Overview | . 6 |
| | 3.3 | Summary of Demographic and Baseline Characteristics | . 7 |
| | 3.4 | Safety Analyses | . 7 |
| | 3.5 | Efficacy Analyses | . 8 |
| | 3.5. | 1 Primary Efficacy Analysis | . 9 |
| | 3.5.2 | 2 Other Efficacy Analyses | 10 |
| | 3.6 | Pharmacokinetic Analyses | 12 |
| 4 | | ple Size Justification | |
| 5 | Inte | rim Analysis | 12 |
| 6 | Gen | neral Information Regarding Data Analyses | 12 |
| 7 | | le Shells | |
| 8 | List | ing Shells | 06 |

#### 1 Introduction

This document provides a description of the statistical methods and procedures to be implemented for the analysis of data from ChemoCentryx, Inc. Protocol CL003\_168. The main purpose of this study was to evaluate the safety and tolerability of CCX168 when given on top on standard of care glucocorticoids and cyclophosphamide or rituximab in patients with antineutrophil cytoplasm antibody (ANCA)-associated vasculitis (AAV). An overview of the study is provided below.

Approximately 45 subjects with AAV were planned to be randomized in a 1:1:1 ratio to one of the following three groups:

Group A: CCX168 10 mg twice daily plus cyclophosphamide/rituximab plus oral corticosteroids;

Group B: CCX168 30 mg twice daily plus cyclophosphamide/rituximab plus oral corticosteroids;

Group C: Placebo twice daily plus cyclophosphamide/rituximab plus oral corticosteroids.

If necessary, rescue corticosteroids can be given to subjects with worsening disease.

Randomization was stratified based on the following three variables:

- Disease status (newly diagnosed AAV or relapsed AAV);
- ANCA positivity (MPO or PR3); and
- Standard of care treatment (cyclophosphamide or rituximab).

Subjects participated in an 84-day treatment period and an 84-day follow-up period. All subjects have scheduled study visits at screening and on Days 1, 2, 8, 15, 22, 29, 43, 57, 71, 85, 99, 113, 141, and 169.

For additional details regarding the study design, please refer to the protocol.

This analysis plan was written after finalization of protocol amendment 4. Any deviations from this analysis plan will be substantiated by sound statistical rationale and documented in the Integrated Clinical and Statistical Report.

### 2 Trial Objectives

The primary safety objective of this study is to evaluate the safety and tolerability of CCX168 in subjects with AAV on background standard of care (SOC) cyclophosphamide or rituximab plus corticosteroid treatment. The primary efficacy objective is to evaluate the efficacy of CCX168 based on the Birmingham Vasculitis Activity Score (BVAS) CCX168 in subjects with AAV on background standard of care cyclophosphamide or rituximab plus corticosteroid treatment.

The secondary objectives of this study include:

- Evaluation of the efficacy of CCX168 plus SOC compared to SOC based on changes in renal disease activity parameters:
  - eGFR (MDRD serum creatinine equation);

- Hematuria (central laboratory microscopic count of urinary RBCs); and
- Albuminuria (first morning urinary albumin:creatinine ratio);
- Assessment of changes in renal inflammatory activity based on urinary monocyte chemoattractant protein-1 (MCP-1):creatinine ratio and serum C-reactive protein (hsCRP) concentration with CCX168 compared to SOC;
- Assessment of health-related quality-of-life changes based on Short Form-36 version 2 (SF-36v2) and EuroQOL-5D-5L (EQ-5D-5L) with CCX168 compared to SOC;
- Assessment of changes in the vasculitis damage index (VDI) with CCX168 compared to SOC;
- Assessment of changes in ANCA (anti-PR3 and anti-MPO) with CCX168 compared to SOC;
- Assessment of changes in pharmacodynamics markers in plasma and urine with CCX168 compared to SOC; and
- Evaluation of the pharmacokinetic profile of CCX168 in subjects with AAV.

### 3 Statistical Methodology

### 3.1 Analysis Populations

For the purposes of data analysis, the intent-to-treat (ITT) Population will include all subjects who are randomized, receive at least one dose of study drug, and have at least one post baseline on-treatment BVAS assessment. Sensitivity analyses will be conducted on the primary efficacy endpoint, disease response, disease remission (BVAS of 0) at Day 85, and disease remission at Day 29 AND 85 including all patients who were randomized. An assessment will be considered to be on treatment if it is observed within 1 day of the last dose of study medication. The safety population will include all subjects who are randomized and receive at least one dose of study drug. A per protocol (PP) population may also be defined if there are major protocol deviations that could affect study outcome.

### 3.2 Analysis Overview

Data will be summarized descriptively by treatment group and overall. For continuous variables, summary statistics will include the sample size, mean, median, standard deviation (SD), standard error of the mean (SEM), minimum, and maximum. Continuous variables with skewed distributions will be log-transformed for analysis including urinary ACR, urinary RBC count, urinary MCP-1:creatinine ratio, and hsCRP. Frequency counts and percentages will be presented for categorical variables. All data will be displayed in data listings which will be included as part of an appendix to the Clinical Study Report.

In analysis tables and listings, the three treatment groups will be referred to as 'Placebo + Standard of Care', 'CCX168 10 mg + Standard of Care', and 'CCX168 30 mg + Standard of Care'. For summaries and analyses for which all subjects randomized to CCX168 treatment are pooled, the treatment group will be referred to as 'All CCX168'.

### 3.3 Summary of Demographic and Baseline Characteristics

All subject baseline characteristics and demographic data (age, sex, race, ethnicity, weight, height, body mass index, smoking status, ECG, TB screen results, viral test results, ANCA, serology test results, vasculitis disease duration (from time of first diagnosis), BVAS, VDI, SF36v2 score, EQ-5D-5L score, hsCRP, eGFR, hematuria, proteinuria (ACR), glomerular histopathology (if biopsy was taken), urinary MCP-1:creatinine ratio, physical examination abnormalities, medical history, previous (within 6 months of screening) and concomitant medications (including vasculitis medication use) at study entry will be listed by treatment group, study center, and subject number, and will also be summarized by treatment group and overall.

### 3.4 Safety Analyses

Safety assessments include adverse events, physical examination abnormalities, vital signs, clinical laboratory tests (including blood chemistry, hematology, and urinalysis), and ECGs.

Safety analyses will be performed on the Safety Population. In general, separate summaries will be prepared for safety events occurring during the 84-day treatment period and the 168-day study period. No inferential analyses will be performed on safety data.

An adverse event will be considered as "pre-treatment" if the start date/time of the event is prior to the time of administration of the first dose of study medication. All other adverse events will be considered "treatment-emergent" (TEAE). Symptoms or signs of vasculitis will be considered adverse events if these increase in severity or frequency while a subject is on study.

An overview of treatment-emergent adverse events will be prepared that presents all TEAEs, serious adverse events (SAEs), TEAEs leading to discontinuation, events related to study medication, corticosteroids, cyclophosphamide, or rituximab, and TEAEs by maximum severity.

Adverse events will be coded using MedDRA and TEAEs will be summarized by system organ class and preferred term. Similar summaries will be prepared for TEAEs related to study medication, corticosteroids, cyclophosphamide, or rituximab, TEAEs by maximum severity, SAEs, and TEAEs leading to discontinuation. Adverse events will be listed by treatment group, including all available information of interest such as onset and resolution dates, study day of onset relative to first dosing day, severity, seriousness, causal relationship to study medication and corticosteroid use, action taken, and outcome.

Laboratory parameter results and changes from baseline will summarized by visit. Shift tables from baseline to subsequent study visits will also be generated. Notable abnormalities will be listed by treatment group and subject number, and will be summarized by treatment group. Laboratory values outside the reference ranges will be flagged in the listings.

Vital sign results and changes from baseline will summarized by visit. Physical examination abnormalities will be summarized by visit and body system. ECG abnormalities will be listed.

The subject incidence of effects possibly associated with glucocorticoid use including serious infections, new-onset diabetes mellitus/hyperglycemia, bone fracture, peptic ulcer disease, cataracts, new onset/worsening hypertension, weight gain more than 10 kg, and psychiatric disorders will be summarized by treatment group for the 84-day treatment period and the 168-day study period. These effects will be identified as follows:

Serious infections: All SAEs in the System Organ Class 'Infections and Infestations'

- New-onset diabetes mellitus/hyperglycemia: All TEAEs of hyperglycemia, diabetes, increased blood glucose, plus all patients with a fasting blood glucose level post-baseline that is above the upper limit of normal on at least two consecutive study visits.
- Bone fracture: All TEAEs indicating long bone or vertebral fractures
- Peptic ulcer disease: All TEAEs indicating upper gastrointestinal ulceration, erosion, or bleeding
- Cataracts: All TEAEs of cataract
- New onset/worsening hypertension: All TEAEs of hypertension, worsening hypertension, or high blood pressure, plus all patients with a systolic blood pressure increase of at least 20 mm Hg from baseline, and >140 mm Hg (systolic), or diastolic blood pressure increase of at least 10 mm Hg from baseline, and >90 mm Hg (diastolic), that is present on at least two consecutive study visits
- Weight gain more than 10 kg: Change from baseline in weight of > 10 kg.
- Psychiatric disorders: All TEAEs of psychosis, anxiety, amnesia, convulsions, delirium, dementia, depression, mania, emotional instability, irritability, euphoria, hallucinations, impaired cognition, increased motor activity, insomnia, memory loss, mania, mood swings, neuritis, neuropathy, paresthesia, personality changes, restlessness, schizophrenia, vertigo, or withdrawal behavior

The subject incidence of infections, serious infections, severe infections (i.e., Grade 3), and infections leading to subject withdrawal from the study will be summarized by treatment group for the 84-day treatment period and the 168-day study period.

### 3.5 Efficacy Analyses

The primary efficacy endpoint is the proportion of subjects achieving disease response at Day 85 defined as BVAS percent reduction from baseline of at least 50% plus no worsening in any body system component.

Other efficacy endpoints include:

- In patients with hematuria and albuminuria at baseline, the proportion of subjects achieving renal response at Day 85; renal response is defined as an improvement in parameters of renal vasculitis:
  - a. an increase from baseline to Day 85 in eGFR (MDRD serum creatinine equation), plus
  - a decrease from baseline to Day 85 in hematuria (central laboratory microscopic count of urinary RBCs), plus
  - a decrease from baseline to Day 85 in albuminuria (first morning urinary albumin:creatinine ratio).
- Proportion of subjects achieving disease remission at Day 85 defined as BVAS of 0;
- Proportion of subjects achieving early disease remission (BVAS of 0) at Day 29 AND Day 85;
- Percent change from baseline to Day 85 in BVAS;
- 5. Change and percent change from baseline to Day 85 in eGFR;

- In subjects with hematuria at baseline (> 5 RBCs/hpf), the percent change from baseline to Day 85 in urinary RBC count;
- In subjects with albuminuria at baseline, the percent change from baseline to Day 85 in urinary ACR;
- 8. Percent change from baseline to Day 85 in urinary MCP-1:creatinine ratio;
- Proportion of subjects requiring rescue glucocorticoid treatment;
- 10. Change from baseline to Day 85 in the VDI;
- Change from baseline to Day 85 in health-related quality-of-life as measured by the SF-36v2 and EQ-5D-5L;

### Other endpoints include:

- Total cumulative study-supplied prednisone dose and duration of dosing during the 84-day treatment period;
- Total cumulative systemic corticosteroid dose (any use) and duration of dosing during the 84-day dosing period;
- Total cumulative cyclophosphamide or rituximab dose and duration of dosing during the 84day dosing period;
- Percent change from baseline in hsCRP;
- 5. Percent change from baseline in ANCA (anti-PR3 and anti-MPO) at Day 85;
- 6. Proportion of patients becoming ANCA negative at Day 85; and
- Change and percent change from baseline in plasma and urine biomarkers.

For all efficacy endpoints, baseline is defined as the last value prior to start of dosing with study medication (typically the Day 1 pre-dose value).

### 3.5.1 Primary Efficacy Analysis

The proportion of subjects achieving disease response (defined above) during the 84-day treatment period will be calculated to compare each CCX168 group against the placebo (standard of care) group. Similar analyses will be performed to compare the All CCX168 group to the placebo group. If the Day 85 result is missing, the last post-randomization result will be used, unless the subject had worsening of AAV and required rescue treatment. In the latter case the subject will be considered a non-responder.

For the purpose of data presentation, the 2-sided 90% confidence intervals will be displayed since the lower bound of the 1-sided 95% confidence interval is identical to the lower bound of the 2-sided 90% confidence interval.

The SAS code used to generate these analyses will be similar to the following:

```
ods listing close;
proc freq data=efficacy order=data;
   tables TRTN*RESP / riskdiff(EQUAL) alpha=0.1;
   weight Frequency;
   ods output RiskDiffCol1=equalc1;
```

```
run;
ods listing;
```

These analyses of disease response will be repeated for the 168-day study period. For this analysis, if the Day 169 result is missing, the last result after Day 85 will be used, unless the subject had worsening of AAV and required rescue treatment. In the latter case the subject will be considered a non-responder.

Subgroup analyses will also be performed for the following subgroups:

- Subjects with renal disease at baseline (defined as subjects with BVAS items scored in the renal organ system)
- Subjects without renal disease at baseline (defined as subjects with no BVAS items scored in the renal organ system)
- 3. Subjects receiving cyclophosphamide background treatment
- 4. Subjects receiving rituximab background treatment
- 5. Subjects with newly diagnosed disease
- 6. Subjects with relapsed disease
- 7. Subjects with MPO+ disease
- 8. Subjects with PR3+ disease
- 9. Subjects with granulomatosis with polyangiitis (Wegener's)
- 10. Subjects with microscopic polyangiitis

For all subgroup analyses, confidence intervals for treatment differences are considered descriptive.

### 3.5.2 Other Efficacy Analyses

Categorical responses will be analyzed using the same approach as the primary efficacy endpoint. This includes:

- Renal response in subjects with hematuria and albuminuria at baseline at Day 85 and at Day 169;
- Disease remission;
- Early disease remission.

Results for subjects who became ANCA negative (PR3 and MPO) at Day 85 and Day 169 will be summarized.

Quantitative efficacy variables will be summarized at each visit as will changes and/or percent changes from baseline. Mixed models for repeated measures (MMRM) will be used to compare treatment groups during the 84-day treatment period and the 168-day study period. Models will include treatment group, visit, treatment-by-visit interaction, AAV disease status (new or

relapsed), ANCA positivity (MPO or PR3), and standard of care treatment (rituximab or cyclophosphamide) as factors and the baseline value as a covariate. The output from the MMRM analysis will include the results at each visit as well as the overall results. P-values from contrasts comparing treatment groups will be presented as will 95% confidence intervals for treatment differences.

Analysis of covariance (ANCOVA) will also be used to compare treatment groups in change and/or percent change from baseline at each visit, for the end of the 84-day treatment period, and the end of the 168-day study period. Models will include AAV disease status (new or relapsed), ANCA positivity (MPO or PR3), and standard of care treatment (rituximab or cyclophosphamide) as factors and the baseline value as a covariate.

The variables to be analyzed in this manner include:

- BVAS percent change from baseline;
- eGFR (MDRD formula) change and percent change from baseline;
- Urinary RBC count ratio and percent change from baseline in subjects with hematuria at baseline;
- ACR ratio and percent change from baseline in subjects with albuminuria at baseline;
- Urinary MCP-1: creatinine ratio and percent change from baseline;
- VDI change and percent change from baseline;
- SF-36 change and percent change from baseline including all domains and the physical component and mental health summaries;
- EQ-5D-5L visual analogue scale and indexed scores change from baseline;
- Serum hsCRP ratio and percent change from baseline;
- ANCA (anti-PR3 and anti-MPO) ratio and percent change from baseline; and
- Serum and urine biomarkers change and percent change from baseline.

The MMRM analyses will be repeated for the BVAS renal subscore and non-renal subscore for the ITT Population only.

Listings of subjects who received rescue treatment will be prepared. Subjects who receive rescue before Day 92 (Day 85 + 7 days) will be considered a treatment failure.

Summaries of dose and duration of study supplied prednisone taken during the 84-day treatment period and the 168-day study period will be provided for the full study population and for each of the subgroups listed above. Similar summaries will be prepared for total systemic corticosteroid treatment, cumulative cyclophosphamide treatment, and cumulative rituximab treatment. A summary of exposure days to randomized treatment (CCX168 or placebo), cumulative CCX168 dose, and percent compliance to the dosing regimen will be provided.

The main efficacy analysis will be in the ITT population. Sensitivity analyses may also be performed excluding subjects with major protocol deviations.

### 3.6 Pharmacokinetic Analyses

The results from pharmacokinetic analyses will be reported in a separate report.

### 4 Sample Size Justification

The sample size was based on practical rather than statistical considerations.

### 5 Interim Analysis

Efficacy and safety data from the study were summarized for review by the DMC at defined points over the course of the study. The DMC charter included details of the analyses.

### 6 General Information Regarding Data Analyses

report for Protocol CL003\_168. All tables and listings will be generated in SAS® version 9.3 or higher and all programs used to generate statistical analyses will be validated according to standard operating procedures. Generally, tables and listings will be printed using Courier New 8pt font with all margins at least one inch. This corresponds to settings in SAS of linesize=134 and pagesize=54. The format of some displays may change slightly depending on the actual length of the data displayed.

# 7 Table Shells

ChemoCentryx, Inc. Protocol CL003 168


Table 14.1.1 Subject Disposition All Enrolled Subjects

Placebo + CCX168 10 mg + CCX168 30 mg + Standard of Care Standard of Care Standard of Care All CCX168 Total Category n (%) n (%) n (%) n (%) n (%)

Screened

Failed screening Reason 1 Reason 2

Randomized

Safety Population

ITT Population

Completed

Early withdrawal on/before Day 85 Subject withdrew consent Sponsor decision Subject lost to follow-up Adverse event Investigator decision Other

Early withdrawal after Day 85 Subject withdrew consent Sponsor decision Subject lost to follow-up Adverse event Investigator decision Other

- Percentage of screen failures is based on the total number of subjects screened. Percentages of Safety population (Intent-to-Treat) population, subjects completed and early withdrawals are based on the number of subjects randomized.

Database last modified: DDMMYYYY Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM

<sup>-</sup> The ITT Population includes all subjects who were randomized and had at least one post baseline on treatment BVAS measurement.

<sup>-</sup> The Safety Population includes all subjects who were randomized and received at least one dose of study drug.


#### Table 14.1.2 Listing of Subjects who Withdrew Prematurely All Randomized Subjects

| Treatment<br>Subject | Age/Sex/Race | Date<br>Randomized | First Dose<br>Date | Withdrawal<br>Date/Day | Last Dose<br>Date/Day | Reason for withdrawal |
|---|---|---|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | #/M/XXXXXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY/## | DDMMMYYYY/## | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | #/M/XXXXXXXXXX | DD <b>MMM</b> YYYY | DD <b>MMM</b> YYYY | DDMMMYYYY/## | DDMMMYYYY/## | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Note: Study day is calculated based on the date of first dose.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYYY

NOTE: This table will be sorted by treatment group and subject within treatment group.

ChemoCentryx, Inc. Protocol CL003\_168


Table 14.1.3 Summary of Subject Demographics All Randomized Subjects

| Demographic Characteristic<br>Statistic/Category | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30 mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) | Total |
|---|---|---|---|---|---|
| Age (Years) | | | | | |
| n | ** | ** | ** | ** | ** |
| Mean | 44.4 | 44.4 | 44.4 | 44.4 | **.* |
| SD | 89.88 | 11.11 | 89.89 | 10.10 | 11.11 |
| SEM | #1.#1 | 11.11 | ##-## | 11.11 | 11.11 |
| Minimum | ** | ** | ** | ** | ** |
| Median | 44.4 | 44.4 | 44.4 | 44.4 | **.* |
| Maximum | ** | ** | ** | ** | ** |
| Gender, n (%) | | | | | |
| Male | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) | ** (***. |
| Female | ## (###.#) | ** (***.*) | ## (###.#) | ** (***.*) | ** (***. |
| Ethnicity, n (%)<br>Hispanic or Latino<br>Not Hispanic or Latino | | | | | |
| Race, n (%) | | | | | |
| Asian | | | | | |
| American Indian or Alaska Native | | | | | |
| Black or African American | | | | | |
| Native Hawaiian or Other | | | | | |
| Pacific Islander | | | | | |
| White | | | | | |
| Other | | | | | |

Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYY Program Name: XXXXXXXX.sas

NOTE: Only non-zero race categories will be included.

#### Table 14.1.4 Summary of Baseline Characteristics All Randomized Subjects

| Baseline Characteristic<br>Statistic/Category | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30 mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) | Total |
|---|---|---|---|---|---|
| Body weight (kg) | | | | | |
| n | ** | ** | ** | ** | ** |
| Mean | 11.1 | 48.4 | 44.4 | 44.4 | 08.0 |
| SD | 11.11 | 99.99 | 11.11 | 11.11 | 98.98 |
| SEM | ##-## | 11.11 | 89.88 | 11.11 | 11.11 |
| Minimum | ** | ** | ** | ** | ** |
| Median | 44.4 | 48.4 | 44.4 | 44.4 | 08.0 |
| Maximum | ** | ** | ** | ** | ** |
| Smoking Status, n (%) | | | | | |
| Current Smoker | ** (***.*) | ## (###-#) | ## (###-#) ## | (###.#) | #0 (0##-#) |
| Past Smoker | | | | | |
| Never Smoked | | | | | |

This table will also include summaries of baseline data for the following parameters:

Height (cm), BMI (kg/m^2), Heart rate, Systolic blood pressure, Diastolic blood pressure, Oral temperature, TB screen results, viral test results, ANCA-newly diagnosed versus relapsed, ANCA associated vasculitis disease duration [1], standard of care (rituximab or cyclophosphamide), anti-MPO+ [2], anti-MPO+ and anti-PR3+ status, type of AAV (GPA, MPO, or renal limited vasculitis), BVAS, VDI, hsCRP, eGFR, hematuria, urine RBC casts, proteinuria (ACR), urinary MCP-1:creatinine ratio, SF-36 domain scores, EQ-5D-5L score and EQ-5D-5L VAS.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY

Note to programmer: For anti-MPO+ and anti-PR3+ status, present the following categories: Only anti-MPO+, Only anti-PR3+, both anti-MPO+ and anti-PR3+, ANCA equivocal, , and both anti-MPO+ and anti-PR3+ negative (see analysese for study CL002\_168).

<sup>[1]</sup> If subject is relapsed, the recorded diagnosis date is used for this summary.

<sup>[2]</sup> For summaries of Anti-MPO+ (IU/mL) and Anti-PR3+ (IU/mL), only subjects with a non-negative baseline categorical status are included. Results reported as '>156.0' are treated as equal to 156.0 for computing summary statistics.

Table 14.1.5 Summary of Prior Medications All Randomized Subjects

| Anatomic Therapeutic Class<br>Preferred Term | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg + Standard of Care (N=##) n (%) | CCX168 30 mg + Standard of Care (N=##) n (%) | All CCX168<br>(N=##)<br>n (%) | Total<br>(N=##)<br>n (%) |
|---|---|---|---|---|---|
| Any Prior Medication | ** (***.*) | ## (###.#) | ** (***.*) | ## (###.#) | ## (###.#) |
| Anatomic Therapeutic Class 1<br>Preferred Term 1 | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) |

<sup>-</sup> Prior medications are defined as any medication taken within 6 months of screening, during the screening period between the screening visit and the day of randomization.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the total column for anatomic therapeutic class and descending frequency in the total column for preferred term within anatomic therapeutic class.

#### Table 14.1.6 Summary of Concomitant Medications All Randomized Subjects

| Anatomic Therapeutic Class<br>Preferred Term | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg +<br>Standard of Care<br>(N=##)<br>n (%) | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | All CCX168<br>(N=##)<br>n (%) | Total<br>(N-##)<br>n (%) |
|---|---|---|---|---|---|
| Any Concomitant Medication | ** (***.*) | ## (###.#) | ** (***.*) | ## (###.#) | ## (###.#) |
| Anatomic Therapeutic Class 1<br>Preferred Term 1 | ** (*#*.#)<br>** (*#*.#) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###-#) |

<sup>-</sup> Concomitant medications are defined as any medication taken on or after the day of randomization.

Frogram Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the total column for anatomic therapeutic class and descending frequency in the total column for preferred term within anatomic therapeutic class.

#### Table 14.1.7.1 Summary of Study Medication Dosing (CCX168/Placebo) All Randomized Subjects

| Dosing Variable | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30 mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|
| Tunation of dosing (days) | | | | |
| Duration of dosing (days) | ** | ** | ** | 44 |
| n<br>Mean | 11.1 | 11.1 | 11.1 | 11.1 |
| SD SD | 11.11 | 11.11 | 11.11 | 11.11 |
| SEM | **.** | **.** | **. ** | **.** |
| Minimum | ***** | **** | *** | ***** |
| Median | 11.1 | 11.1 | 11.1 | 11.1 |
| Maximum | *** | ** | ** | ** |
| MORINGE | ** | ** | ** | ** |
| Total CCX168 Dose (mg)* | | | | |
| n | ** | ** | ** | ** |
| Mean | 44.4 | 88.8 | 44.4 | **.* |
| SD | 44.44 | 44.44 | 40.40 | 44.44 |
| SEM | ##.## | 11.11 | ##.## | 11.11 |
| Minimum | ** | ** | ** | ** |
| Median | 44.4 | 44.4 | 44.4 | **.* |
| Maximum | ** | ** | ** | ** |
| Overall Percent Compliance | | | | |
| n | ** | ** | ** | ** |
| Mean | 11.1 | 11.1 | **.* | 11.1 |
| SD | **.** | **.** | **.** | **.** |
| SEM | 44.44 | 44.44 | 80.80 | 66.66 |
| Minimum | ** | ** | ** | ** |
| Median | **.* | **.* | **.* | **.* |
| Maximum | 44 | 44 | 44 | 6.6 |

<sup>\*</sup>Subjects who did not return any capsules of study medication at last day of 84-dosing period will be excluded from total dose and overall compliance calculation.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYY HH:MM

Note to programmer: Duration of dosing—date of last dose – date of first dose + 1. Total CCX168 dose=0 for subjets randomized to placebo; =number of capsules taken\*10/3 for subjects randomized to CCX168 10 mg + SOC; =number of capsules taken\*10 for subjects randomized to CCX168 30 mg + SOC.

# The following table will have the same layout as Table 14.1.7.1:

Table 14.1.7.2 Summary of Study Medication Dosing (CCX168/Placebo) Intent-to-Treat Population

#### Table 14.2.1.1 Analysis of BVAS Response Intent-to-Treat Population

| Day | Treatment | N' | n | (8) | Difference<br>in percentages<br>versus Placebo | Two-sided 90% CI<br>for Difference |
|---|---|---|---|---|---|---|
| Day 85 | Placebo + Standard of Care (N=##) CCX168 10 mg + Standard of Care (N=##) CCX168 30 mg + Standard of Care (N=##) All CCX168 (N=##) | *** | *** | (###.#)<br>(###.#)<br>(###.#)<br>(###.#) | **.**<br>**.**<br>**.** | (#.##, #.##)<br>(#.##, #.##)<br>(#.##, #.##) |
| epeat for | Day 169 | | | | | |

Repeat for Day 169

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYY

<sup>-</sup> BVAS response is defined as achieving a 50% reduction from baseline in the BVAS plus no worsening in any body system component.

N = number of subjects in the analysis population for the specified treatment group; N'=number of subjects with post-baseline on treatment BVAS data; n=number of responders; %=100\*n/N'

### The following tables will have the same layout as Table 14.2.1.1:

Table 14.2.1.2

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.1.3

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.1.4

Analysis of BVAS Response

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.1.5

Analysis of BVAS Response

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.1.6

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.1.7

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.1.8

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.1.9

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.1.10

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.1.11

Analysis of BVAS Response

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Table 14.2.1.12

Analysis of BVAS Response

All Randomized Patients


#### Table 14.2.2.1 Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population

| Day | Treatment | N' | n | (3) | Difference<br>in percentages<br>versus Placebo | Two-sided 90% CI<br>for Difference |
|---|---|---|---|---|---|---|
| Day 85 | Placebo + Standard of Care (N=##) CCX168 10 mg + Standard of Care (N=##) CCX168 30 mg + Standard of Care (N=##) All CCX168 (N=##) | *** | *** | (###.#)<br>(###.#)<br>(###.#)<br>(###.#) | #*.#*<br>#*.#*<br>#*.#* | (#.##, #.##)<br>(#.##, #.##)<br>(#.##, #.##) |

Repeat for Day 169

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYY

<sup>-</sup> Renal response at Day 85 is defined as improvement in the following parameters of renal vasculitis: (1) increase from baseline to Day 85 in eGFR (MDRD equation), (2) decrease from baseline to Day 85 in hematuria (microscopic count of urinary RBCs), and decrease from baseline to Day 85 in albuminuria (first morning urinary albumin; creatinine ratio).

<sup>-</sup> N = number of subjects in the analysis population for the specified treatment group; N'=number of subjects with post-baseline BVAS data; n=number of responders; %=100\*n/N'

### The following tables will have the same layout as Table 14.2.2.1:

#### Table 14.2.2.2

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

#### Table 14.2.2.3

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

#### Table 14.2.2.4

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

#### Table 14.2.2.5

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

#### Table 14.2.2.6

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

#### Table 14.2.2.7

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

#### Table 14.2.2.8

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

#### Table 14.2.2.9

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

#### Table 14.2.2.10

Analysis of Renal Response for Patients with Hematuria and Albuminuria at Baseline
All Randomized Patients

#### Table 14.2.3.1 Analysis of BVAS Disease Remission Intent-to-Treat Population

| Day | Treatment | N' | n | (8) | Difference<br>in percentages<br>versus Placebo | Two-sided 90% CI<br>for Difference |
|---|---|---|---|---|---|---|
| Day 85 | Placebo + Standard of Care (N=##) CCX168 10 mg + Standard of Care (N=##) CCX168 30 mg + Standard of Care (N=##) All CCX168 (N=##) | *** | *** | (###.#)<br>(###.#)<br>(###.#)<br>(###.#) | ##.##<br>##.##<br>##.## | (#.##, #.##)<br>(#.##, #.##)<br>(#.##, #.##) |

Repeat for Day 169

- Disease remission is defined as achieving a BVAS score of 0. Subjects with missing data have the last observation carried forward.

Frogram Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYYY

<sup>-</sup> N = number of subjects in the analysis population for the specified treatment group; N'=number of subjects with post-baseline on treatment BVAS data; n=number of responders; %=100\*n/N'

### The following tables will have the ame layout as Table 14.2.3.1:

Table 14.2.3.2

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.3.3

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.3.4

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.3.5

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.3.6

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.3.7

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.3.8

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.3.9

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.3.10

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.3.11

Analysis of BVAS Disease Remission

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Table 14.2.3.12

Analysis of BVAS Disease Remission

All Randomized Patients

# Table 14.2.4.1 Analysis of Early Disease Remission Intent-to-Treat Population

| Treatment | N' | n | (%) | Difference<br>in percentages<br>versus Placebo | Two-sided 90% CI<br>for Difference |
|---|---|---|---|---|---|
| Placebo + Standard of Care (N=##) CCX168 10 mg + Standard of Care (N=##) CCX168 30 mg + Standard of Care (N=##) All CCX168 (N=##) | *** | *** | (###.#)<br>(###.#)<br>(###.#)<br>(###.#) | #*.##<br>#*.## | (*.#*, *.#*)<br>(*.#*, *.#*)<br>(*.#*, *.#*) |

<sup>-</sup> Early disease remission is defined as achieving a BVAS score of 0 at Day 29 and Day 85. Subjects with missing data at either Day 29 or Day 85 are considered to not have achieved early disease remission.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYYY

<sup>-</sup> N = number of subjects in the analysis population for the specified treatment group; N'=number of subjects with post-baseline on treatment BVAS data; n=number of responders; %=100\*n/N'

### The following tables will have the ame layout as Table 14.2.4.1:

Table 14.2.4.2

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.4.3

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.4.4

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.4.5

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.4.6

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.4.7

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.4.8

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.4.9

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.4.10

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.4.11

Analysis of Early Disease Remission

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Table 14.2.4.12

Analysis of Early Disease Remission

All Randomized Patients


Table 14.2.5.1 Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population

| Study Day<br>Statistic | Placebo +<br>Standard of Care<br>(N=##) | | CCX168 10 mg +<br>Standard of Care<br>(N=##) | | CCX168 30 mg +<br>Standard of Care<br>(N=##) | | All CCX168<br>(N=##) | |
|---|---|---|---|---|---|---|---|---|
| | Visit | % Change | Visit | % Change | Visit | % Change | Visit | % Change |
| Baseline | | | | | | | | |
| N' | ** . | | | | | | | |
| Mean<br>SD | **.** | | | | | | | |
| SEM | 44.44 | | | | | | | |
| Minimum | ** | | | | | | | |
| Median | **.* | | | | | | | |
| Maximum | ** | | | | | | | |
| Day 29 | | | | | | | | |
| N' | 44 | ## | ** | 8.0 | 4.6 | ## | 6.6 | 0.6 |
| Mean | 46.4 | 44.4 | 48.4 | ##.# | 48.4 | 80.8 | **.* | 46.4 |
| SD | **-** | ##-## | **-** | ##-## | **-** | ##-## | 11.11 | **-** |
| SEM<br>Minimum | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Median | 11.1 | 11.1 | 11.1 | 11.1 | 11.1 | 11.1 | 11.1 | 11.1 |
| Maximum | ** | ** | ** | ** | ** | ## | ** | ** |
| P-value* | | | | 4.4444 | | 4.4444 | | 4.4444 |
| 95% CI* | | | | (-##.#, ##.#) | | (-##.#, ##.#) | | (-#0.#, #0. |

<sup>-</sup> Baseline is defined as the last pre-dose value.

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from a MMRM model with treatment group, visit, treatment-by visit interaction, AAV disease status (new or relapsed), and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate.

ChemoCentryx, Inc. Protocol CL003 168


Table 14.2.5.1 Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population

| Study Day<br>Statistic | Placebo + Standard of Care (N=##) | | CCX168 10 mg +<br>Standard of Care<br>(N=##) | | CCX168 30 mg +<br>Standard of Care<br>(N=##) | | All CCX168<br>(N=##) | |
|---|---|---|---|---|---|---|---|---|
| | Visit | % Change | Visit | % Change | Visit | % Change | Visit | % Change |
| Day 85 | | | | | | | | |
| N' | ** | ** . | ** | ** . | ** . | ** . | ** . | ** |
| Mean | **.* | **.* | **.* | **.* | **.* | **.* | **.*. | **.*. |
| SD<br>SEM | 11.11 | 11.11 | 11.11 | 80.80<br>81.81 | 99.00 | 44.44<br>41.41 | 11.11 | 11.11 |
| Minimum | ** | ** | ** | ** | ** | ** | ** | ** |
| Median | **.* | 11.1 | **.* | 11.1 | **.* | 11.1 | **.* | **.* |
| Maximum | ** | ** | ** | ## | *** | ## | ** | 0.0 |
| P-value* | | | | +. ++++ | | +. ++++ | | *.**** |
| 95% CI* | | | ( | (-##.#, ##.#) | | (-##.#, ##.#) | | (-#0.#, #0. |
| Overall | | | | | | | | |
| N' | ** | ** | ** | ** | ** | ** | ** | ** |
| Mean | 44.4 | **.* | 44.4 | ##.# | 44.4 | ##.# | **.* | **.* |
| SD | **-** | **-** | **-** | **-** | **-** | **-** | 11.11 | **-** |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum<br>Median | 11.1 | 11.1 | ** | ## # | 11.1 | ## # | 11.1 | *** |
| Maximum | *** | ## | *** | ## | *** | *** | *** | 98.7 |
| P-value* | ** | ** | ** | +. ++++ | ** | *.**** | ** | *.**** |
| 95% CI* | | | | (-##.#, ##.#) | | (-##.#, ##.#) | | (-#0.#, #0. |

<sup>-</sup> Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

Note to programmer: For summary statistics in the 'Overall' category, first calculate the average value for a subject then combine subjects to obtain summary statistics.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from a MMRM model with treatment group, visit, treatment-by visit interaction, AAV disease status (new or relapsed), and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate.

### The following tables will have the a similar layout as Table 14.2.5.1:

#### Table 14.2.5.2

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Renal Disease at Baseline

#### Table 14.2.5.3

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

#### Table 14.2.5.4

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

#### Table 14.2.5.5

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

#### Table 14.2.5.6

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

#### Table 14.2.5.7

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Relapsed Disease

#### Table 14.2.5.8

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with MPO+ Disease

#### Table 14.2.5.9

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with PR3+ Disease

#### Table 14.2.5.10

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

#### Table 14.2.5.11

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis Table 14.2.5.12

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients

Table 14.2.5.13

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.5.14

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.5.15

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.5.16

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.5.17

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.5.18

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.5.19

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.5.20

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.5.21

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.5.22

Summary and Analysis (MMRM) of BVAS Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Note to programmer: The MMRM tables for the 168-day study period will include summaries for each post-baseline visit and the p-value and 95% confidence interval for the overall differences between each group and placebo. This comment applies to all MMRM tables for the 168-day study period.

### The tables below will have the same layout as Tables 14.2.5.1 and 14.2.5.12:

#### Table 14.2.5.23

Summary and Analysis (MMRM) of BVAS Renal Sub-score Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population

#### Table 14.2.5.24

Summary and Analysis (MMRM) of BVAS Renal Sub-score Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population

#### Table 14.2.5.25

Summary and Analysis (MMRM) of BVAS Non-renal Sub-score Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population

#### Table 14.2.5.26

Summary and Analysis (MMRM) of BVAS Non-renal Sub-score Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population

# Table 14.2.5.27 Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population

| Study Day<br>Statistic | Placebo +<br>Standard of Care<br>(N=##) | | CCX168 10 mg + Standard of Care (N=##) | | CCX168 30 mg +<br>Standard of Care<br>(N=##) | | All CCX168<br>(N=##) | |
|---|---|---|---|---|---|---|---|---|
| | Visit | % Change | Visit | % Change | Visit | % Change | Visit | % Change |
| Baseline | | | | | | | | |
| N' | ** | | | | | | | |
| Mean | **-* | | | | | | | |
| SD | **.** | | | | | | | |
| SEM<br>Minimum | **.** | | | | | | | |
| Median | **.* | | | | | | | |
| Maximum | ** | | | | | | | |
| Day 29 | | | | | | | | |
| N' | ** | ## | 4.6 | ## | 4.6 | ## | 6.6 | 0.6 |
| Mean | 44.4 | 80.8 | 48.4 | **.* | 48.4 | 44.4 | **.* | **.* |
| SD | **-** | #1.## | **-** | **-** | **-** | **-** | 11.11 | **-** |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum<br>Median | ** | ** . | ** . | ** . | ** . | ** . | ** . | ** . |
| Maximum | ** | #1.1 | **-* | ##.# | **-* | ## . # | ** | **-* |
| P-value* | *** | ** | ** | 4.4444 | ** | 4.4444 | ** | 4.4444 |
| 95% CI* | | | | (-##.#, ##.#) | | (-##.#, ##.#) | | (-#0.#, #0.0 |

The additional visits to be summarized include:

Day 85, End of Treatment, Day 113, Day 169, End of Follow-up

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from ANCOVA models with treatment group, AAV disease status (new or relapsed) and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate.

### The following tables will have the same layout as Table 14.2.5.27:

Table 14.2.5.28

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.5.29

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.5.30

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline
Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.5.31

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.5.32

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.5.33

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.5.34

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.5.35

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.5.36

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.5.37

Summary and Analysis (ANCOVA) of BVAS Percent Change from Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis
ChemoCentryx, Inc. Protocol CL003 168


Table 14.2.6.1 Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population

| | Sta | Placebo +<br>ndard of<br>(N=##) | | Sta | X168 10 mg<br>ndard of (<br>(N=##) | Care | | X168 30mg<br>ndard of<br>(N=##) | | A | 11 CCX168<br>(N=##) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day<br>Statistic | Visit | Change | % Change | Visit | Change | % Change | Visit | Change | | Visit | Change | % Chang |
| Baseline | | | | | | | | | | | | |
| N' | ** | | | | | | | | | | | |
| Mean | **.** | | | | | | | | | | | |
| SD | **.*** | | | | | | | | | | | |
| SEM<br>Minimum | **.* | | | | | | | | | | | |
| Median | **.** | | | | | | | | | | | |
| Maximum | 11.1 | | | | | | | | | | | |
| Day 2 | | | | | | | | | | | | |
| N' | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | 40 | #0 |
| Mean | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | ##-## |
| SD | **.** | **.** | **.*** | **.** | **.*** | **.*** | **.** | **.*** | **.*** | **.*** | **.** | **.*** |
| SEM<br>Minimum | 98.888 | **.** | **.** | **.** | 11.1 | 11.1 | **.** | **.** | **.* | ##.### | 10.1 | 10.1 |
| Median | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Maximum | 46.4 | 44.4 | 44.4 | 44.4 | 44.4 | 44.4 | 44.4 | 44.4 | **.* | | 40.4 | 40.4 |
| P-value* | | | | | | 1.0000 | | | 1.0110 | | | 1.1111 |
| 95% CI for C | | | | | (-##-#, | | | (-##-#, | ##-#) | | (-##.#, | 0f.0) |
| 95% CI for % | Change* | | | | (-##.#, # | <b>##.#</b> ) | | (-##.#, | ##.#) | | (-##.#, | ##.#) |

The additional visits to be summarized include:

Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, and Overall

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from a MMRM model with treatment group, visit, treatment-by visit interaction, AAV disease status (new or relapsed), and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate.

# The following tables will have layout similar to Table 14.2.6.1:

#### Table 14.2.6.2

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with Renal Disease at Baseline

### Table 14.2.6.3

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

#### Table 14.2.6.4

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

## Table 14.2.6.5

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

### Table 14.2.6.6

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

# Table 14.2.6.7

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Relapsed Disease

### Table 14.2.6.8

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.6.9

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with PR3+ Disease

# Table 14.2.6.10

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

### Table 14.2.6.11

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population

## Table 14.2.6.13

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Renal Disease at Baseline

## Table 14.2.6.14

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

# Table 14.2.6.15

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

### Table 14.2.6.16

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.6.17

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Fercent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

## Table 14.2.6.18

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Relapsed Disease

## Table 14.2.6.19

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.6.20

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with PR3+ Disease

### Table 14.2.6.21

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

### Table 14.2.6.22

Summary and Analysis (MMRM) of eGFR (MDRD) Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis Page 1 of #

Table 14.2.6.23 Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population

| Study Day | Sta | Placebo +<br>ndard of<br>(N=##) | Care | Sta | x168 10 mg<br>ndard of (<br>(N=##) | Care | Sta | X168 30mg<br>ndard of<br>(N=##) | Care | | All CCX1 | 1) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day<br>Statistic | Visit | Change | % Change | Visit | Change | % Change | Visit | Change | % Change | Visit | | & Change |
| Baseline | | | | | | | | | | | | |
| N' | ** | | | | | | | | | | | |
| Mean | 11.11 | | | | | | | | | | | |
| SD | **.*** | | | | | | | | | | | |
| SEM | **.** | | | | | | | | | | | |
| Minimum | 99.9 | | | | | | | | | | | |
| Median | **.** | | | | | | | | | | | |
| Maximum | **.* | | | | | | | | | | | |
| Day 2 | | | | | | | | | | | | |
| N' | ** | ** | ** | ** | ** | 4.6 | ** | ** | 44 | ** | 40 | 40 |
| Mean | **.** | **.** | **.** | **.** | **.** | **.** | **.** | 80.80 | 80.80 | 80.80 | **.** | 80.80 |
| SD | 99.999 | **-*** | **.*** | **-*** | **-*** | **-*** | **.** | **.** | **.** | **.** | **.** | **-** |
| SEM | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** |
| Minimum | 46.4 | 46.4 | 46.4 | **.* | **.* | 46.4 | 80.6 | 80.8 | 80.8 | 80.8 | 40.4 | 40.4 |
| Median | **-** | **-** | **.** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** | **-** |
| Maximum | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* |
| P-value* | | | | | | | | | 4.0000 | | | *. **** |
| 95% CI for C | | | | | (-##-#, 1 | | | (-##-#, | | | (-##.#, | |
| 95% CI for % | Change* | | | | (-##.#, 1 | †#-#) | | (-##-#, | ##-#) | | (-##.#, | 0f.0) |

The additional visits to be summarized include:

Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, End of Treatment, Day 99, Day 113, Day 141, Day 169, and End of Follow-up Period.

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from ANCOVA models with treatment group, AAV disease status (new or relapsed) and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate.

# The following tables will have the same layout as Table 14.2.6.23:

### Table 14.2.6.24

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

#### Table 14.2.6.25

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

#### Table 14.2.6.26

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

## Table 14.2.6.27

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.6.28

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

## Table 14.2.6.29

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

### Table 14.2.6.30

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.6.31

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

# Table 14.2.6.32

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

## Table 14.2.6.33

Summary and Analysis (ANCOVA) of eGFR (MDRD) Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis ChemoCentryx, Inc. Protocol CL003 168


Table 14.2.7.1 Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Hematuria at Baseline

| Shorter Sans | | Placebo mard of (N=##) | | | X168 10 m<br>ndard of (<br>(N=##) | | | X168 30mg<br>ndard of<br>(N=##) | | All CCX168<br>(N=##) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day<br>Statistic | Visit | Ratio | % Change | Visit | Ratio | & Change | Visit | Ratio % | Change | Visit | Ratio | & Chang |
| Baseline<br>N'<br>Mean<br>Geo. Mean (GM)<br>Minimum<br>Median<br>Maximum | ## | | | | | | | | | | | |
| ay 2<br>N'<br>Mean<br>Geo. Mean (GM)<br>Minimum<br>Median<br>Maximum<br>P-value^<br>95% CI^ for Rat | **<br>**.**<br>**.**<br>**.**<br>**.* | **<br>**.**<br>**.**<br>**.** | **<br>**.**<br>**.** | ##<br>##.##<br>##.##<br>##.##<br>##.# | **<br>**.**<br>**.**<br>**.**<br>**.** | **.** | | ##<br>##.##<br>##.##<br>##.##<br>##.## | ##<br>##.##<br>##.##<br>##.## | | #0<br>#0.#0<br>#0.#0<br>#0.#0<br>#0.#0<br>#0.#0 | ##<br>##.#<br>##.# |

Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, and Overall

Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> Ratio is defined for each subject as the visit value divided by the baseline value.

<sup>\*</sup> Since urinary-RBC values are reported as ranges, quantitative values are defined as: 75 for result of '>75', 50 for '50-75', 30 for '30-49', 16 for '16-29', 10 for '10-15', 6 for '6-9', 3 for '3-5', 1 for '1-2', 0.5 for 'occ', and 0.1 for 'None'.

<sup>^</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from a MMRM model with treatment group, visit, treatment-by visit interaction, AAV disease status (new or relapsed), and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate. Logarithmic transformations were applied to the data before fitting the ANCOVA model. The 95% confidence interval was transformed back to the original scale.

# The following tables will a layout similar Table 14.2.7.1:

#### Table 14.2.7.2

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Hematuria at Baseline and Receiving Cyclophosphamide Background Treatment

# Table 14.2.7.3

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Fatients with Hematuria at Baseline and Receiving Rituximab Background Treatment

#### Table 14.2.7.4

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Newly Diagnosed Disease

## Table 14.2.7.5

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - Patients with Hematuria at Baseline and Relapsed Disease

### Table 14.2.7.6

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Hematuria at Baseline and MPO+ Disease

## Table 14.2.7.7

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Hematuria at Baseline and PR3+ Disease

### Table 14.2.7.8

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Hematuria at Baseline and Granulomatosis Polyangiitis (Wegener's)

# Table 14.2.7.9

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Microscopic Polyangiitis

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Steps 1 through 3 Combined

Intent-to-Treat Population - Patients with Hematuria at Baseline

#### Table 14.2.7.11

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Hematuria at Baseline and Receiving Cyclophosphamide Background Treatment

#### Table 14.2.7.12

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Receiving Rituximab Background Treatment

## Table 14.2.7.13

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Fercent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Hematuria at Baseline and Newly Diagnosed Disease

#### Table 14.2.7.14

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Relapsed Disease

## Table 14.2.7.15

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and MPO+ Disease

#### Table 14.2.7.16

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and PR3+ Disease

#### Table 14.2.7.17

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Polyangiitis (Wegener's)

## Table 14.2.7.18

Summary and Analysis (MMRM) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Hematuria at Baseline and Microscopic Polyangiitis


Table 14.2.7.19 Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline

| | | Placebo : ndard of (N=##) | | | X168 10 :<br>ndard of<br>(N=##) | Care | | X168 30m<br>indard of<br>(N=##) | | A. | All CCX168<br>(N=##) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day<br>Statistic | Visit | Ratio | % Change | Visit | Ratio | % Change | Visit | Ratio | t Change | Visit | Ratio | & Change |
| Baseline | | | | | | | | | | | | |
| N' | ** | | | | | | | | | | | |
| Mean | **-** | | | | | | | | | | | |
| Geo. Mean (GM) | **.** | | | | | | | | | | | |
| Minimum<br>Median | **.* | | | | | | | | | | | |
| Maximum | **.* | | | | | | | | | | | |
| Day 2<br>N' | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| Mean | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Geo. Mean (GM) | **.*** | 44.444 | ***** | 44.444 | 40.000 | ***** | 44.444 | 44.444 | **.** | 44.444 | **.** | **.** |
| Minimum | **.* | **.* | **.* | **-* | 11.1 | **.* | ** ** | ##.# | **.* | **.* | 10.1 | **.* |
| Median | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Maximum | **.* | 44.4 | 44.4 | 44.4 | 44.4 | 48.4 | 80.6 | 80.8 | 44.4 | 44.4 | 40.4 | 40.4 |
| P-value^ | | | | | 0.0000 | | | | | | | |
| 95% CI^ for Rat | io | | | (-# | .**, *.* | #) | (-#. | **, *.** | ) | (-#. | **, *.**) | |

Additional visits to be summarized include:

Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, End of Treatment, Day 99, Day 113, Day 141, Day 169, and End of Follow-up Period.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

<sup>-</sup> Ratio is defined for each subject as the visit value divided by the baseline value.

<sup>\*</sup> Since urinary-RBC values are reported as ranges, quantitative values are defined as: 75 for result of '>75', 50 for '50-75', 30 for '30-49', 16 for '16-29', 10 for '10-15', 6 for '6-9', 3 for '3-5', 1 for '1-2', 0.5 for 'Occ', and 0.1 for 'None'.

<sup>^</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from ANCOVA models with treatment group, AAV disease status (new or relapsed), and ANCA positivity (MPO or PR3) as factors and the baseline value as a covariate. Logarithmic transformations were applied to the data before fitting the ANCOVA model. The 95% confidence interval was transformed back to the original scale.

# The following tables will have the same layout as Table 14.2.7.19:

### Table 14.2.7.20

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population - Patients with Hematuria at Baseline and Receiving Cyclophosphamide Background Treatment

## Table 14.2.7.21

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and Receiving Rituximab Background Treatment

## Table 14.2.7.22

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and Newly Diagnosed Disease

## Table 14.2.7.23

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and Relapsed Disease

## Table 14.2.7.24

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and MPO+ Disease

# Table 14.2.7.25

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and PR3+ Disease

### Table 14.2.7.26

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and Granulomatosis with Polyangiitis (Wegener's)

# Table 14.2.7.27

Summary and Analysis (ANCOVA) of Urinary RBC\* Count: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Hematuria at Baseline and Microscopic Polyangiitis

# The following tables will have layouts similar to to Tables 14.2.7.x

#### Table 14.2.8.1

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline

### Table 14.2.8.2

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Cyclophosphamide Background Treatment

# Table 14.2.8.3

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Rituximab Background Treatment

## Table 14.2.8.4

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline and Newly Diagnosed Disease

## Table 14.2.8.5

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Relapsed Disease

## Table 14.2.8.6

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and MPO+ Disease

### Table 14.2.8.7

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and PR3+ Disease

# Table 14.2.8.8

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Granulomatosis Polyangiitis (Wegener's)

# Table 14.2.8.9

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Microscopic Polyangiitis

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline

#### Table 14.2.8.11

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Cyclophosphamide Background Treatment

## Table 14.2.8.12

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Rituximab Background Treatment

# Table 14.2.8.13

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline and Newly Diagnosed Disease

### Table 14.2.8.14

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline and Relapsed Disease

## Table 14.2.8.15

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline and MPO+ Disease

## Table 14.2.8.16

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 160-day Study Period
Intent-to-Treat Population - Patients with Albuminuria at Baseline and PR3+ Disease

### Table 14.2.8.17

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Polyangiitis (Wegener's)

### Table 14.2.8.18

Summary and Analysis (MMRM) of ACR: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - Patients with Albuminuria at Baseline and Microscopic Polyangiitis

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline

## Table 14.2.8.20

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Cyclophosphamide Background Treatment

## Table 14.2.8.21

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population - Patients with Albuminuria at Baseline and Receiving Rituximab Background Treatment

#### Table 14.2.8.22

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and Newly Diagnosed Disease

### Table 14.2.8.23

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and Relapsed Disease

## Table 14.2.8.24

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and MPO+ Disease

## Table 14.2.8.25

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and PR3+ Disease

## Table 14.2.8.26

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population - Patients with Albuminuria at Baseline and with Granulomatosis Polyangiitis (Wegener's)

### Table 14.2.8.27

Summary and Analysis (ANCOVA) of ACR: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - Patients with Albuminuria at Baseline and Microscopic Polyangiitis

# The following tables will have layouts similar to to Tables 14.2.7.x

Table 14.2.9.1

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population

Table 14.2.9.2

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.9.3

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.9.4

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.9.5

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.9.6

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.9.7

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.9.8

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with MPO+ Disease

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with PR3+ Disease

## Table 14.2.9.10

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Granulomatosis Polyangiitis (Wegener's)

# Table 14.2.9.11

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population

Table 14.2.9.13

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.9.14

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.9.15

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.9.16

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.9.17

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.9.18

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.9.19

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with MPO+ Disease

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with PR3+ Disease

## Table 14.2.9.21

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Granulomatosis Polyangiitis (Wegener's)

# Table 14.2.9.22

Summary and Analysis (MMRM) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population

#### Table 14.2.9.24

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

## Table 14.2.9.25

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

#### Table 14.2.9.26

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

### Table 14.2.9.27

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

# Table 14.2.9.28

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

## Table 14.2.9.29

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population - All Patients with Relapsed Disease

### Table 14.2.9.30

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.9.31

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

### Table 14.2.9.32

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Granulomatosis Polyangiitis (Wegener's)

### Table 14.2.9.33

Summary and Analysis (ANCOVA) of Urinary MCP-1:Creatinine Ratio: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis ChemoCentryx, Inc. Protocol CL003\_168


# Table 14.2.10.1 Listing of Rescue Glucocorticoid Treatment Intent-to-Treat Population

RT: Reported Term

Treatment ATC: Anatomic Therapeutic Class Start Date (Day) / Duration

Subject PT: Preferred Term End Date (Day) Dose/Unit Route/Frequency Indication (Days)

DDMMMYYYY (###)/ ## XXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXX 

DDMMMYYYY (###)

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM ChemoCentryx, Inc. Protocol CL003\_168


# Table 14.2.10.2 Listing of All Systemic Glucocorticoid Treatment Intent-to-Treat Population

RT: Reported Term

Treatment ATC: Anatomic Therapeutic Class Start Date (Day) / Duration

Subject PT: Preferred Term End Date (Day) Dose/Unit Route/Frequency Indication (Days)

Program Name: XXXXXXXX.sas

DDMMMYYYY (###)/ ## XXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXX 

DDMMMYYYY (###)

Database last modified: DDMMYYYY HH:MM

Run Date: DDMMMYYYY HH:MM

# The following tables will have similar layouts to Tables 14.2.5.x:

#### Table 14.2.11.1

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population

#### Table 14.2.11.2

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Renal Disease at Baseline

#### Table 14.2.11.3

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

## Table 14.2.11.4

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

### Table 14.2.11.5

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.11.6

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

### Table 14.2.11.7

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Relapsed Disease

# Table 14.2.11.8

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.11.9

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with PR3+ Disease

### Table 14.2.11.10

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

## Table 14.2.11.11

Summary and Analysis (MMRM) of VDI Change and Percent Change from Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis Table 14.2.11.12

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population

Table 14.2.11.13

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.11.14

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.11.15

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.11.16

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.11.17

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.11.18

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.11.19

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.11.20

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.11.21

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.11.22

Summary and Analysis (ANCOVA) of VDI Change and Percent Change from Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis Page 1 of #

# Table 14.2.12.1 Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population

CCV160 30mg +

CCV168 10 mg +

| Domain<br>Study Day | | Placebo +<br>ndard of<br>(N=##) | | | x168 10 m<br>ndard of<br>(N=##) | | | x168 30mg<br>indard of<br>(N=##) | | | All CCX16<br>(N=##) | 8 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Statistic | Visit | Change | % Change | Visit | Change | % Change | Visit | Change | % Change | Visit | Change | & Change |
| Physical Funct | ioning | | | | | | | | | | | |
| Baseline<br>N' | | | | | | | | | | | | |
| Mean | **.** | | | | | | | | | | | |
| SD | 44.444 | | | | | | | | | | | |
| SEM | 11.111 | | | | | | | | | | | |
| Minimum | **.* | | | | | | | | | | | |
| Median | 48.48 | | | | | | | | | | | |
| Maximum | 99.9 | | | | | | | | | | | |
| Day 29 | | | | | | | | | | | | |
| n' | 44 | 4.6 | 4.6 | ** | ** | 4.6 | ** | ** | 44 | 44 | 40 | 40 |
| Mean | 99.99 | 99.99 | **.** | 99.99 | **.** | **.** | **.** | 89.89 | 89.89 | **.** | 89.89 | 89.80 |
| SD | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.*** | **.** | **.*** | **.*** | **.*** | **.*** |
| SEM | **.*** | **.*** | **.*** | 48.466 | **.** | **.** | **.** | **.** | **.** | **.** | 80.805 | 44.406 |
| Minimum | **.* | **.* | **.* | **-* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | 10.1 |
| Median | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Maximum | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | **.* | 40.4 | 40.4 |
| P-value* | | | | | 1.1111 | 1.1111 | | 1.1111 | 1.1111 | | 1.1111 | 1.1111 |
| 95% CI for C | | | | | (-##.#, | | | | ##-#) | | (-##.#, | |
| 95% CI for % | change* | | | | (-##.#, | ##·#) | | (-##.#, | *#.*) | | (-##.#, | **-*) |

The domains to be summarized include:

Role-Physical, Role-Emotional, Social Functioning, Bodily Pain, Mental Health, Vitality, General Health Perceptions, Change in Health, Physical Component Summary, Mental Health Summary.

The additional visits to be summarized include: Day 29, Day 85, End of Treatment, Day 169, and End of Follow-up Period.

placabo +

Program Name: XXXXXXXX.sas Database last modified: DDMMYYYY HH:MM Run Date: DDMMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

<sup>\*</sup>P-values and 95% confidence intervals for differences between specified treatment groups and placebo are from a MMRM model with treatment group as a factor and randomization strata (AAV status, ANCA positivity, and standard of care treatment) as covariates.

# The following table will have similar layouts to Tables 14.2.12.1:

Table 14.2.12.2

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.12.3

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.12.4

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.12.5

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.12.6

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.12.7

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.12.8

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.12.9

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.12.10

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.12.11

Summary of SF-36 v2.0: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

# The following table will have similar layouts to Tables 14.2.12.1:

#### Table 14.2.13.1

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit
Intent-to-Treat Population

#### Table 14.2.13.2

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit
Intent-to-Treat Population - All Patients with Renal Disease at Baseline

#### Table 14.2.13.3

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit
Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

## Table 14.2.13.4

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

## Table 14.2.13.5

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.13.6

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

### Table 14.2.13.7

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Relapsed Disease

# Table 14.2.13.8

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit
Intent-to-Treat Population - All Patients with MPO+ Disease

# Table 14.2.13.9

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with PR3+ Disease

### Table 14.2.13.10

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

## Table 14.2.13.11

Summary of EQ-5D-5L Health Scale Score and VAS: Actual, Change and Percent Change from Baseline by Visit Intent-to-Treat Population - All Patients with Microscopic Polyangiitis 

# Table 14.2.14 Summary of Dose and Duration of Study Supplied Prednisone Intent-to-Treat Population

| Ad-day treatment period, N' (%) ## (###.#) ## (###.#) ## (###.#) Total study-supplied prednisone/placebo dose (mg) N' Mean SD SEM Minimum Median Median Maximum | Period<br>Variable | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|---|
| N' Mean SD SEM Minimum Median | 4-day treatment period | , N' (%) ## (###-#) | ## (###-#) | ## (###-#) | ** (***.*) |
| Mean SD SEM Minimum Median | | prednisone/placebo dose (m | ng) | | |
| SD<br>SEM<br>Minimum<br>Median | | | | | |
| SEM<br>Minimum<br>Median | | | | | |
| Minimum<br>Median | | | | | |
| Median | | | | | |
| | Maximum | | | | |
| | | dy-supplied predmisone/pla | (days) | | |
| Total duration of study-supplied prednisone/placebo use (days) | | | | | |
| N' | SD | | | | |
| N'<br>Mean | SEM | | | | |
| N' Mean SD | Minimum | | | | |
| N' Mean SD SEM | Median | | | | |
| N' Mean SD SEM Minimum | Maximum | | | | |

<sup>-</sup> N' = number of subjects who took study supplied prednisone during the designated study period.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY 

# Table 14.2.15 Summary of Dose and Duration of Total Systemic Corticosteroid Treatment\* Intent-to-Treat Population

| Period<br>Variable | Placebo + Standard of Care (N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|
| 84-day treatment period, N' (% | ) ## (###-#) | ## (###-#) | ## (###-#) | ## (###.#) |
| Total systemic corticostero | id dose (mg) | | | |

Mean

SD

SEM

Minimum

Median Maximum

Total duration of systemic corticosteroid use (days)

N'

Mean

SD

SEM

Minimum

Median

Maximum

Repeat for 168-day study period

Database last modified: DDMMYYYY Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM

<sup>-</sup> N' = number of subjects who took corticosteroid during the designated study period.

<sup>\*</sup>Total systemic (IV and oral) corticosteroid treatment includes (1) study-supplied prednisone use, (2) new corticosteroid use, and (3) maintenance corticosteroid use over the course of the trial.


# Table 14.2.16.1 Summary of Total Cumulative Cyclophosphamide Dose Intent-to-Treat Population

| Period<br>Variable | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|
| 84-day treatment period, N' (% | ) ## (###·#) | ## (###-#) | ## (###-#) | ** (***.*) |
| Total cumulative dose (mg) | | | | |
| N' | | | | |
| Mean | | | | |
| SD | | | | |
| SD | | | | |
| SEM<br>Minimum | | | | |
| Median | | | | |
| Maximum | | | | |
| manal durantian of desire (d | | | | |
| Total duration of dosing (do | ays) | | | |
| Mean | | | | |
| SD | | | | |
| SEM | | | | |
| Minimum | | | | |
| Median | | | | |
| Maximum | | | | |

Repeat for 168-day study period

Program Name: XXXXXXXX.sas Database last modified: DDMMYYYY Run Date: DDMMMYYYY HH:MM

<sup>-</sup> N' = number of subjects who took at least one dose of cyclophosphamide during the designated study period.

<sup>-</sup> Cyclophosphamide dose was calculated as recorded amount (mg/kg) \*weight at that visit. If weight was missing, the last weight for that subject would be used.

ChemoCentryx, Inc. Protocol CL003\_168


# Table 14.2.16.2 Summary of Total Cumulative Rituximab Dose Intent-to-Treat Population

| Period<br>Variable | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30mg + Standard of Care (N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|
| 84-day treatment period, N' | (%) ## (###.#) | ## (###-#) | ## (###-#) | ** (***.*) |

Total cumulative dose (mg)

Mean

SD

SEM

Minimum

Median

Maximum

Total duration of dosing (days)

Mean SD

SEM

Minimum

Median

Maximum

Repeat for 168-day study period

- N' = number of subjects who took at least one dose of cyclophosphamide during the designated study period.

Program Name: XXXXXXXX.sas Database last modified: DDMMYYYY Run Date: DDMMMYYYY HH:MM

The following tables will have similar layouts to Tables 14.2.7.x:

(For these tables, the last footnote will be '- Results of '< 0.2' were imputed to have a value of 0.2 for analysis.')

## Table 14.2.17.1

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population

### Table 14.2.17.2

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Renal Disease at Baseline

### Table 14.2.17.3

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

## Table 14.2.17.4

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

## Table 14.2.17.5

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.17.6

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

### Table 14.2.17.7

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Relapsed Disease

## Table 14.2.17.8

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with MPO+ Disease

## Table 14.2.17.9

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with PR3+ Disease

# Table 14.2.17.10

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

## Table 14.2.17.11

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period
Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

## Table 14.2.17.12

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population

# Table 14.2.17.13

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Renal Disease at Baseline

## Table 14.2.17.14

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

# Table 14.2.17.15

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Treatment Period
Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

### Table 14.2.17.16

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

## Table 14.2.17.17

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

## Table 14.2.17.18

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Relapsed Disease

## Table 14.2.17.19

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with MPO+ Disease

### Table 14.2.17.20

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with PR3+ Disease

### Table 14.2.17.21

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period
Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

### Table 14.2.17.22

Summary and Analysis (MMRM) of Serum hsCRP: Ratio and Percent Change Compared to Baseline during the 168-day Study Period Intent-to-Treat Population - All Patients with Microscopic Polyangiitis Table 14.2.17.23

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population

Table 14.2.17.24

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.17.25

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.17.26

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.17.27

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.17.28

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.17.29

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.17.30

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.17.31

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.17.32

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Steps 1 through 3 Combined

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.17.33

Summary and Analysis (ANCOVA) of Serum hsCRP: Ratio and Percent Change Compared to Baseline Steps 1 through 3 Combined

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

# The following tables will have similar layouts to Tables 14.2.7.x:

Table 14.2.18.1

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population

Table 14.2.18.2

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.18.3

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 94-day Treatment Period

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.18.4

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.18.5

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 94-day Treatment Period

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.18.6

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.18.7

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 94-day Treatment Period

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.18.8

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MP0): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with MPO+ Disease

## Table 14.2.18.9

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with PR3+ Disease

## Table 14.2.18.10

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

# Table 14.2.18.11

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 84-day Treatment Period

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

Table 14.2.18.12

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population

Table 14.2.18.13

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.18.14

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.18.15

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.18.16

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.18.17

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.18.18

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.18.19

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with MPO+ Disease

## Table 14.2.18.20

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with PR3+ Disease

## Table 14.2.18.21

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

# Table 14.2.18.22

Summary and Analysis (MMRM) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline during the 168-day Study Period

Intent-to-Treat Population - All Patients with Microscopic Polyangiitis
Table 14.2.18.23

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population

Table 14.2.18.24

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.18.25

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.18.26

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.18.27

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.18.28

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline
Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.18.29

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.18.30

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with MPO+ Disease

Table 14.2.18.31

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with PR3+ Disease

Table 14.2.18.32

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.18.33

Summary and Analysis (ANCOVA) of ANCA (anti-PR3 and anti-MPO): Ratio and Percent Change Compared to Baseline Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

## Table 14.2.19.1 Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population

| Parameter<br>Day | Treatment | N' | n | (%) | Difference<br>in percentages<br>versus Placebo |
|---|---|---|---|---|---|
| R3 (cANCA) | antibody by ELISA | | | | |
| Day 85 | Placebo + Standard of Care (N=##) CCX168 10 mg + Standard of Care (N=##) CCX168 30 mg + Standard of Care (N=##) All CCX168 (N=##) | *** | *** | (###.#)<br>(###.#)<br>(###.#) | ***.*<br>***.* |
| epeat for | Day 169 | | | | |
| epeat for | parameter: MPO (pANCA) antibody by ELISA | (IU/mL) | | | |

<sup>-</sup> N'=number of subjects who were PR3 positive (for PR3 analysis) and MPO positive (for MPO analysis) at baseline with post-baseline ANCA data during the specified dosing period.

Program Name: XXXXXXXX.sas Database last modified: DDMMYYYY Run Date: DDMMMYYYY HH:MM

## The following tables will have the ame layout as Table 14.2.19.1:

Table 14.2.19.2

Analysis of Subjects who Became ANCA Negative
Intent-to-Treat Population - All Patients with Renal Disease at Baseline

Table 14.2.19.3

Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population - All Patients with Non-Renal Disease at Baseline

Table 14.2.19.4

Analysis of Subjects who Became ANCA Negative
Intent-to-Treat Population - All Patients Receiving Cyclophosphamide Background Treatment

Table 14.2.19.5

Analysis of Subjects who Became ANCA Negative
Intent-to-Treat Population - All Patients Receiving Rituximab Background Treatment

Table 14.2.19.6

Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population - All Patients with Newly Diagnosed Disease

Table 14.2.19.7

Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population - All Patients with Relapsed Disease

Table 14.2.19.8

Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population - All Patients with Granulomatosis with Polyangiitis (Wegener's)

Table 14.2.19.9

Analysis of Subjects who Became ANCA Negative Intent-to-Treat Population - All Patients with Microscopic Polyangiitis

## Table 14.3.1.1 Overview of Treatment-emergent Adverse Events during the 84-day Treatment Period Safety Population

| cebo + CCX168 10 mg + CCX168 30 mg + rd of Care Standard of Care Standard of Care All CCX16 |
|---|
| -##) (N-##) (N-##) (N-##)<br>(%) n (%) n (%) n (%) |
| (***.*) |
| _ |

Mild Moderate Severe Life-threatening

#### Serious TEAE

Possibly-Study Medication Related Serious TEAE Possibly-Corticosteroid Use Related Serious TEAE Possibly-Cyclophosphamide Related Serious TEAE Possibly Azathioprine Related Serious TEAE Possibly Rituximab Related Serious TEAE

#### Discontinued study medication due to TEAE

Due to Possibly-Study Medication Related Serious TEAE

Due to Possibly-Corticosteroid Use Related TEAE

Due to Possibly-Corticosteroid Use Related Serious TEAE

Due to Possibly-Cyclophosphamide Related TEAE

Due to Possibly-Cyclophosphamide Related Serious TEAE

Due to Possibly-Rituximab Related TEAE

Due to Possibly- Rituximab Related Serious TEAE

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

## The following tables will have the same layout as Table 14.3.1.1:

Table 14.3.1.2 Overview of Treatment-emergent Adverse Events during the 168-day Study Period Safety Population


#### Table 14.3.1.3 Summary of Treatment-emergent Adverse Events During the 94-Day Treatment Period by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg + Standard of Care (N=##) n (%) | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | All CCX168<br>(N=##)<br>n (%) |
|---|---|---|---|---|
| Any Treatment-emergent Adverse Event | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| System Organ Class 1<br>Preferred Term 1 | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#) | ## (###.#) |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

## The following table will have the same layout as Table 14.3.1.3:

Table 14.3.1.4

Summary of Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class and Preferred Term

Safety Population

Table 14.3.1.5 Summary of Treatment-emergent Adverse Events during the 168-day Treament Period by System Organ Class, Preferred Term and Relationship to Study Drug Safety Population

| System Organ Class<br>Preferred Term | Placebo +<br>Standard of Care<br>(N=##) | CCX168 10 mg +<br>Standard of Care<br>(N=##) | CCX168 30 mg +<br>Standard of Care<br>(N=##) | All CCX168<br>(N=##) |
|---|---|---|---|---|
| Relationship to Study Drug | n (%) | n (%) | n (%) | n (%) |
| Any Treatment-emergent Adverse Event | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Possibly related to study drug | ## (###.#) | ## (###.#) | ## (###.#) | 0# (##0.#) |
| Probably not related to study drug | ## (###-#) | ## (###-#) | ## (###-#) | ** (***.*) |
| System Organ Class 1 | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Possibly related to study drug | ## (###-#) | ## (###-#) | ## (###-#) | 0f (ff0.f) |
| Probably not related to study drug | ** (***.*) | ** (***.*) | ** (***.*) | ** (***.*) |
| Preferred Term 1 | ## (###.#) | ## (###-#) | ## (###-#) | 08 (880.8) |
| Possibly related to study drug | ## (###.#) | ## (###.#) | ## (###.#) | ** (***.*) |
| Probably not related to study drug | ## (###.#) | ## (###.#) | ## (###.#) | 0# (##0.#) |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

CL003 168

Table 14.3.1.6

Summary of Treatment-emergent Adverse Events during the 84-day Treatment Period by System Organ Class, Preferred Term and Relationship to Corticosteroid Use Safety Population

| System Organ Class Preferred Term Relationship to Corticosteroid Use | Placebo +<br>Standard of Care<br>(N=##)<br>n (%) | | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | All CCX168<br>(N=##)<br>n (%) |
|---|---|---|---|---|
| Overall | N-## | N-## | N-## | N=## |
| Any Treatment-emergent Adverse Event | ## (###-#) | ## (###-#) | ** (***.*) | ## (###-#) |
| Possibly related to corticosteroid use | ## (###-#) | ## (###-#) | ## (###-#) | ## (###.#) |
| Probably not related to corticosteroid use | ## (###.#) | ## (###.#) | ** (***.*) | ## (###.#) |
| System Organ Class 1 | ## (###.#) | ## (###.#) | ## (###.#) | ** (***.*) |
| Possibly related to corticosteroid use | ## (###.#) | ## (###.#) | ** (***.*) | ## (###.#) |
| Probably not related to corticosteroid use | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Preferred Term 1 | ** (***.*) | ## (###.#) | ## (###.#) | ** (***.*) |
| Possibly related to corticosteroid use | ## (###.#) | ## (###.#) | ## (###.#) | 0# (##0.#) |
| Probably not related to corticosteroid use | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Frogram Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

## The following table will have the same layout as Table 14.3.1.6:

## Table 14.3.1.7

Summary of Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class, Preferred Term and Relationship to Corticosteroid Use Safety Population

Table 14.3.1.8

Summary of Treatment-emergent Adverse Events during the 84-day Treatment Period by System Organ Class, Preferred Term and Relationship to Cyclophosphamide Use Safety Population

| System Organ Class Preferred Term | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg +<br>Standard of Care<br>(N=##)<br>n (%) | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | (N=##) |
|---|---|---|---|---|
| Relationship to Cyclophosphamide Use | ц (е) | п (е) | п (е) | n (%) |
| Any Treatment-emergent Adverse Event | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Possibly related to cyclophosphamide use | ## (###-#) | ** (***.*) | ## (###-#) | ## (###.#) |
| Probably not related to cyclophosphamide use | ## (###-#) | ** (***-*) | ## (###-#) | ## (###-#) |
| system Organ Class 1 | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Possibly related to cyclophosphamide use | ## (###.#) | ** (***.*) | ## (###-#) | ** (***-*) |
| Probably not related to cyclophosphamide use | ** (***.*) | ** (***.*) | ** (***.*) | ** (***.*) |
| Preferred Term 1 | ** (***.*) | ** (***.*) | ## (###-#) | ** (***-*) |
| Possibly related to cyclophosphamide use | ** (***.*) | ** (***.*) | ** (***.*) | ** (***.*) |
| Probably not related to cyclophosphamide use | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |

An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

## The following table will have the same layout as Table 14.3.1.8:

## Table 14.3.1.9

Summary of Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class, Preferred Term and Relationship to Cyclophosphamide Use Safety Population

# Table 14.3.1.10 Summary of Treatment-emergent Adverse Events during the 84-day Treatment Period by System Organ Class, Preferred Term and Relationship to Rituximab Use Safety Population

| System Organ Class<br>Preferred Term<br>Relationship to Rituximab Use | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg + Standard of Care (N=##) n (%) | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | All CCX168<br>(N=##)<br>n (%) |
|---|---|---|---|---|
| Any Treatment-emergent Adverse Event Possibly related to rituximab use Probably not related to rituximab use | ## (###.#)<br>## (###.#) | 00 (000.0)<br>00 (000.0)<br>00 (000.0) | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#)<br>## (###.#) |
| System Organ Class 1 Possibly related to rituximab use Probably not related to rituximab use | ** (***.*) | ** (***.*) | ## (###.#) | ## (###.#) |
| | ** (***.*) | ** (***.*) | ## (###.#) | ## (###.#) |
| | ** (***.*) | ** (***.*) | ## (###.#) | ## (###.#) |
| Preferred Term 1 | ** (***.*) | ** (***.*) | ## (###.#) | ## (###.#) |
| Possibly related to rituximab use | ** (***.*) | ** (***.*) | ## (###.#) | ## (###.#) |
| Probably not related to rituximab use | ** (**.*) | ** (**.*) | ## (###.#) | ## (###.#) |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Frogram Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

## The following table will have the same layout as Table 14.3.1.10:

## Table 14.3.1.11

Summary of Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class, Preferred Term and Relationship to Rituximab Use Safety Population


Table 14.3.1.12 Summary of Treatment-emergent Adverse Events during the 94-day Treatment Period by System Organ Class, Preferred Term and Maximum Severity Safety Population

| | Placebo + | CCX168 10 mg + | CCX168 30 mg + | |
|---|---|---|---|---|
| System Organ Class | Standard of Care | Standard of Care | Standard of Care | All CCX168 |
| Preferred Term | (N=##) | (N=##) | (N=##) | (N=##) |
| Maximum Severity | n (%) | n (%) | n (%) | n (%) |
| Any Treatment-emergent Adverse Event | ** (***.*) | ## (###.#) | ## (###.#) | ## (###.#) |
| Mild | ## (###.#) | ** (***.*) | *# (##*-#) | ** (***-*) |
| Moderate | ## (###-#) | ** (***.*) | *# (##*-#) | ** (***-*) |
| Severe | ** (***.*) | ** (***.*) | ** (***.*) | ** (***.*) |
| Life-threatening | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Death | ## (###-#) | ** (***-*) | ** (***-*) | ** (***-*) |
| System Organ Class 1 | ## (###.#) | ## (###.#) | ## (###.#) | |
| Mild | ## (###·#) | ** (***.*) | ## (###-#) | ## (###-#) |
| Moderate | ** (***.*) | ** (***.*) | ** (***.*) | ** (***.*) |
| Severe | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Life-threatening | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Death | ## (###-#) | ## (###-#) | ## (###-#) | ** (***-*) |
| Preferred Term 1 | ## (###.#) | ## (###.#) | ## (###.#) | |
| Mild | ## (###·#) | ** (***.*) | ## (###-#) | ## (###-#) |
| Moderate | ## (###.#) | ** (***.*) | ** (***.*) | ** (***.*) |
| Severe | ## (###.#) | ** (***.*) | ## (###.#) | ## (###.#) |
| Life-threatening | ## (###-#) | ## (###-#) | ## (###-#) | ## (###-#) |
| Death | ## (###-#) | ** (***.*) | ## (###-#) | ## (###.#) |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM

NOTE: Table will be sorted by descending frequency in the All CCX168 column for system organ class and preferred term within system organ class.

NOTE: If there are no events in a category, e.g. Death, the row will not appear in the summary table.

## The following table will have the same layout as Table 14.3.1.12:

Table 14.3.1.13

Summary of Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class, Preferred Term and Maximum Severity Safety Population


Table 14.3.1.14 Summary of Treatment-emergent Adverse Effects Possibly Associated with Glucocorticoid Use during the 84-day Treatment Period by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Placebo + Standard of Care (N=##) n (%) | CCX168 10 mg + Standard of Care (N=##) n (%) | CCX168 30 mg +<br>Standard of Care<br>(N=##)<br>n (%) | All CCX168<br>(N=##)<br>n (%) |
|---|---|---|---|---|
| Any Treatment-emergent Adverse Effect | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.#) |
| Serious Infections<br>New onset diabetes/hyperglycemia | ## (###.#)<br>## (###.#) | ## (###-#)<br>## (###-#) | ** (*#*.#)<br>** (*#*.#) | ## (###.#)<br>## (###.#) |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

## Note to Programmer: These adverse effects will be identified as follows:

- Serious infections: All SAEs in the System Organ Class Infections and Infestations
- New-onset diabetes mellitus/hyperglycemia: All TEAEs of hyperglycemia, diabetes, increased blood glucose, plus all patients with a fasting blood glucose level post baseline that is above the upper limit of normal on at least two consecutive study visits.
- Bone fracture: All TEAEs indicating long bone or vertebral fractures
- Peptic ulcer disease: All TEAEs indicating upper gastrointestinal ulceration, erosion, or bleeding
- Cataracts: All TEAEs of cataract
- New onset/worsening hypertension: All TEAEs of hypertension, worsening hypertension, or high blood pressure, plus all patients with a systolic blood pressure increase of at least 20 mm Hg from baseline, and >140 mm Hg (systolic), or diastolic blood pressure increase of at least 10 mm Hg from baseline, and >90 mm Hg (diastolic), that is present on at least two consecutive study visits.
- Weight gain more than 10 kg: Change from baseline in weight of > 10 kg.
- Psychiatric disorders: All TEAEs of psychosis, anxiety, amnesia, convulsions, delirium, dementia, depression, mania, emotional instability, irritability, euphoria, hallucinations, impaired cognition, increased motor activity, insomnia, memory loss, mania, mood swings, neuritis, neuropathy, paresthesia, personality changes, restlessness, schizophrenia, vertigo, or withdrawal behavior.

## The following table will have the same layout as Table 14.3.1.14:

Table 14.3.1.15

Summary of Treatment-emergent Adverse Effects Possibly Associated with Glucocorticoid Use during the 168-day Study Period by System Organ Class and Preferred Term

Safety Population

#### Table 14.3.1.16 Summary of Treatment-emergent Infections\* during the 84-day Treatment Period by System Organ Class and Preferred Term Safety Population

| | Placebo + | CCX168 10 mg + | CCX168 30 mg + | N11 00916 |
|---|---|---|---|---|
| Sustan Organ Class | Standard of Care | Standard of Care | Standard of Care | All CCX16 |
| System Organ Class | (N=##) | (N=##) | (N=##) | (N=##) |
| Preferred Term | n (%) | n (%) | n (%) | n (%) |
| Any Treatment-emergent Infection | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.# |
| Any Serious Treatment-emergent Infection | ## (###.#) | ## (###.#) | ## (###.#) | ## (###.# |
| Any Severe Treatment-emergent Infection | ** (***.*) | ## (###-#) | ## (###-#) | ## (###-# |
| Any Treatment-emergent Infection Leading to Withdrawal | ** (***.*) | ** (***.*) | ## (###.#) | ** (***.* |
| System Organ Class 1 | ** (***.*) | ## (###-#) | ## (###-#) | ## (###.# |
| Preferred Term 1 | ## (###.#) | ** (***.*) | ## (###.#) | ## (###.# |

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>\*</sup>Summary table includes treatment-emergent infections including serious infections, severe infections (i.e., Grade 3), and infections Leading to withdrawal from the study.

## The following table will have the same layout as Table 14.3.1.16:

Table 14.3.1.17

Summary of Treatment-emergent Infections\* during the 168-day Study Period by System Organ Class and Preferred Term

Safety Population

## The following tables will have the same layouts as Tables in Section 14.3.1:

Table 14.3.1.18

Summary of Serious Treatment-emergent Adverse Events during the 84-Day Treatment Period by System Organ Class and Preferred Term Safety Population

Table 14.3.1.19

Summary of Serious Treatment-emergent Adverse Events during the 168-day Study Period by System Organ Class and Preferred Term Safety Population

Table 14.3.1.20

Summary of Treatment-emergent Adverse Events Leading to Discontinuation of Study Medication Safety Population


#### Table 14.3.2.1 Listing of Serious Adverse Events Safety Population

RT: Reported Term ----- SAE -----Treatment OC: Primary System Organ Class Start Date (Day)/ Related- Action Out-Improve/ Reappear/ Subject TEAE? PT: Preferred Term End Date (Day) Severity ness[1] Taken[2] come[3,4] Disappear[5] Worsen[6] \*\*\*-\*\*\* DDMMYYYY (###) / XXXXXXXX #/#/# XX DDMMMYYYY (###) OC:XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX Last Dose Date (Day): DDMMYYYYY (###) Cumulative Dose (mg) [7]:###

- [1] Relatedness: (Study Medication/Corticosteroid/Cyclophosphamide) 0=Probably Not Related, 1=Possibly Related
- [2] Actions Taken: 1=None, 2=Study medication discontinued, 3=Study medication interrupted
- [3] Outcome: 1=Resolved, 2=Resolved with seguelae, 3=Ongoing, 4=Death, 5=Unknown
- [4] Serious Cutcome: 1=Results in death, 2=Life threatening, 3=Inpatient hospitalization or prolongation of existing hospitalization, 4=Persistent or significant disability/incapacity, 5=Congenital abnormality or birth defect, 6=Important medical event
- [5] Did the event improve or disappear after stopping study medication (dechallenge)?
- [6] Did the event reappear or worsen after restarting study medication (rechallenge)?
- [7] Represents the cumulative dose (mg) of CCX168 taken prior to onset of event.

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM

NOTE: This table will be sorted by treatment group and subject within treatment group.

NOTE: Cumulative dose for placebo subjects will be 0 mg.

<sup>-</sup> An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication. 'Day' is the number of days from the date of randomization.

## The following table will have the same layout as Table 14.3.2.1:

Table 14.3.2.2 Listing of Adverse Events Leading to Discontinuation of Study Medication Safety Population

> Table 14.3.2.3 Listing of Treatment-emergent Infections Safety Population

## Table 14.3.4.1 Summary of Changes in Hematology Laboratory Parameters by Visit Safety Population

| Parameter<br>Study Day<br>Statistic | | ebo +<br>d of Care<br>##)<br>Change | Standar | 10 mg +<br>d of Care<br>##)<br>Change | | 30 mg +<br>d of Care<br>##)<br>Change | All<br>(N= | CCX168<br>##)<br>Change |
|---|---|---|---|---|---|---|---|---|
| Parameter 1 (U<br>Baseline | Init) | | | | | | | |
| N' | ** | | ** | | ** | | ** | |
| Mean | 11.1 | | **.* | | **.* | | 11.1 | |
| SD | **.** | | **.** | | **.** | | **.** | |
| SEM | 48.48 | | 44.44 | | 44.44 | | 44.44 | |
| Minimum | ** | | ** | | ** | | ** | |
| Median | **.* | | **.* | | **.* | | **.* | |
| Maximum | ** | | ** | | ** | | ** | |
| Day 2 | | | | | | | | |
| N' | 44 | ** | ** | 84 | ** | ** | ** | 0.6 |
| Mean | 44.4 | 80.8 | **.* | 80.8 | **.* | 80.8 | **.* | **.* |
| SD | **-** | **-** | **-** | **-** | 11.11 | ##-## | 11.11 | 11.11 |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum | ** | ** | ** | ** | ** | ** | ** | ** |
| Median | 11.1 | ##.# | **-* | ##-# | 11.1 | ##-# | **** | **-* |
| Maximum | ** | ** | ** | ** | ** | ** | ** | ** |

The laboratory parameters to be summarized include:

Hematology: Hematocrit, RBC Count, WBC Count (with both absolute and % differential), Platelet count, MCH, MCHC and MCV.

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 29, Day 43, Day 71, Day 85, End of Treatment, Day 99, Day 141, Day 169, End of Follow-up Period.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

#### Table 14.3.4.2 Summary of Changes in Chemistry Laboratory Parameters by Visit Safety Population

| Parameter<br>Study Day<br>Statistic | udy Day (N=##) | | CCX168 10 mg + Standard of Care (N=##) Visit Change | | CCX168 30 mg + Standard of Care (N=##) Visit Change | | All CCX168<br>(N=##)<br>Visit Change | |
|---|---|---|---|---|---|---|---|---|
| Parameter 1 (U | Jnit) | | | | | | | |
| Baseline | | | | | | | | |
| N' | ** | | ** | | ** | | ** | |
| Mean | **-* | | **-* | | **.* | | **** | |
| SD | **.** | | **.** | | **.** | | **.** | |
| SEM | **.** | | **.** | | **.** | | **.** | |
| Minimum | ** | | ** | | ** | | ** | |
| Median | **.* | | **.* | | **.* | | **.* | |
| Maximum | ** | | ** | | ** | | ** | |
| Day 2 | | | | | | | | |
| N' | 4.6 | ## | ** | ** | ** | ** | 44 | 0.6 |
| Mean | **.* | 80.8 | 44.4 | ##.# | 44.4 | 80.8 | 44.4 | 44.4 |
| SD | **.** | ##.## | **.** | ##.## | **.** | ##.## | 11.11 | **.** |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum | ** | ## | ** | ## | ** | ## | 6.6 | 0.6 |
| Median | **.* | **.* | **-* | **.* | **.* | **.* | 11.1 | **-* |
| Maximum | ** | ** | ** | ** | ** | ** | ** | ** |

The laboratory parameters to be summarized include:

Total Bilirubin, LDH, SGOT/AST, SGPT/ALT, BUN, Creatinine, CPK, Albumin, Sodium, Potassium, Bicarbonate, Chloride, Calcium, Inorganic phosphorus, Glucose, Total protein, Alkaline phosphatase, Cholesterol and Uric acid.

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 29, Day 43, Day 71, Day 85, End of Treatment, Day 99, Day 141, Day 169, End of Follow-up Period.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

## Table 14.3.4.3 Summary of Changes in Urinalysis Laboratory Parameters by Visit Safety Population

| Parameter | Standar | ebo +<br>d of Care | Standar | 10 mg +<br>d of Care | | d of Care | | CCX168 |
|---|---|---|---|---|---|---|---|---|
| Study Day<br>Statistic | Visit (N= | ##)<br>Change | Visit | ##)<br>Change | Visit (N= | f#)<br>Change | Visit (N= | Change |
| Parameter 1 (U | nit) | | | | | | | |
| Baseline | | | | | | | | |
| N' | ** . | | ** . | | ** . | | !! . | |
| Mean<br>SD | **-* | | **-* | | **-* | | 11.1 | |
| SEM | **.** | | **.** | | **.** | | **.** | |
| Minimum | ***** | | *** | | ***** | | ***** | |
| Median | | | **.* | | **.* | | **.* | |
| Maximum | **.* | | **** | | **** | | *** | |
| PRATITION | ** | | ** | | ** | | ** | |
| Day 2 | | | | | | | | |
| N' | ** | 8.0 | ** | 8.0 | 44 | 8.0 | 6.6 | 0.6 |
| Mean | 48.4 | 44.4 | 44.4 | 44.4 | 44.4 | 44.4 | 44.4 | 46.0 |
| SD | 11.11 | **.** | **-** | **.** | **-** | **.** | 11.11 | 11.11 |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum | 4.6 | ## | 4.6 | 84 | 4.6 | ** | 6.6 | 0.6 |
| Median | **-* | **.* | **-* | **.* | **-* | **.* | 11.1 | 08.0 |
| Maximum | ** | ** | ** | ** | ** | ** | ** | ** |

The laboratory parameters to be summarized include: pH and specific gravity.

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 29, Day 43, Day 71, Day 85, End of Treatment, Day 99, Day 141, Day 169, End of Follow-up Period.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

## Table 14.3.4.4 Shift Table for Categorical Changes in Hematology Parameters by Visit Safety Population

| Davamatar/Normal Dangal | Visit | Trastmant | Baseline | | at Specified | |
|---|---|---|---|---|---|---|
| Parameter (Normal Range) | VISIC | Treatment | Category | <lian< th=""><th>NOTHAL</th><th>&gt;ULN</th></lian<> | NOTHAL | >ULN |
| Parameter 1 (###-###) | Day 2 | Placebo+Standard of Care (N'=## ) | < LLN<br>Normal<br>> ULN | ## (###.#)<br>## (###.#) | ## (###.#)<br>## (###.#) | ## (###.#<br>## (###.# |
| | | CCX168 10 mg+Standard of Care (N'=# | <b>#</b> ) | | | |
| | | CCX168 10 mg+Standard of Care (N'=# | <b>#</b> ) | | | |
| | | All CCX168 (N'=##) | | | | |

The laboratory parameters to be summarized will include:

Hemoglobin, Hematocrit, Red blood cell count, White blood cell count (with differential), Platelet count, MCH, MCHC and MCV.

Chemistry: Total Bilirubin, LDH, SGOT/AST, SGPT/ALT, BUN, Creatinine, CPK, Albumin, Sodium, Potassium, Bicarbonate, Chloride, Calcium, Inorganic phosphorous, Glucose, Total protein, Alkaline phosphatase, Cholesterol, and Uric acid.

Urinalysis: pH and specific gravity.

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 29, Day 43, Day 71, Day 85, End of Treatment, Day 99, Day 141, Day 169, End of Follow-up Period.

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM

<sup>-</sup> N'= number of subjects in group with assessment of parameter at baseline and specified visit

<sup>-</sup> n = number of subjects in group with post-baseline measurement outside specified limit

<sup>- % = 100\*</sup>n/N'

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

The following table will have the same layout as Table 14.3.4.4:

Table 14.3.4.5
Shift Table for Categorical Changes in Chemistry Parameters by Visit
Safety Population

The parameters to be summarized in Table 14.3.4.5 include: Total Bilirubin, LDH, SGOT/AST, SGPT/ALT, BUN, Creatinine, CPK, Albumin, Sodium, Potassium, Bicarbonate, Chloride, Calcium, Inorganic phosphorous, Glucose, Total protein, Alkaline phosphatase, Cholesterol, and Uric acid.

## Table 14.3.4.6 Shift Table for Categorical Urinalysis Parameters by Visit Safety Population

| Parameter<br>Visit | Baseline<br>Value | Post-<br>Baseline<br>Value | Placebo +<br>Standard of Care<br>n (%) | CCX168+<br>Standard of Care<br>n (%) | CCX168+<br>Standard of Care<br>n (%) | All CCX168 |
|---|---|---|---|---|---|---|
| Parameter 1 | | | N'-## | N'-## | N'-## | N'-## |
| Day 2 | Category 1 | Category 1<br>Category 2<br>Category n | ** (***.*) | ** (***.*) | ## (###.#) | ** (***.*) |

The urinalysis parameters include:

Glucose, Nitrite, Ketones, Bilirubin, Blood Urobilinogen, RBC, and WBC

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, End of Treatment, Day 99, Day 113, Day 141, Day 169, End of Follow-up Period.

- N'= number of subjects in group with baseline and post-baseline measurements of specified parameter
- n = number of subjects in group with post-baseline measurement outside specified limit
- % = 100\*n/N'
- The End of Treatment value is the last measurement through Day 85.
- The End of Follow-up Period is the last measurement after Day 85 through Day 169.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM


## Table 14.3.4.6 Listing of Laboratory Data for Subjects with Notable Laboratory Abnormalities Safety Population

| Treatment<br>Subject Parameter (Unit) | Normal<br>Range | Visit (Study Day) | Value | Clinical<br>Significance |
|---|---|---|---|---|
| ***** | xxxx-xxxx | XXXXXXXXXXXXXX (##) | *********** | NOTABLE HIGH |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY

NOTE: The table will include all records for each parameter that has at least one occurrence of a NOTABLE or CRITICAL abnormality as identified by the central laboratory. This table will be sorted by treatment group and subject within treatment group.

#### Table 14.3.5.1 Summary of Changes in Vital Signs, Weight, and BMI by Visit Safety Population

| Parameter<br>Study Day<br>Statistic | | ebo +<br>d of Care<br>##)<br>Change | Standar | 10 mg +<br>d of Care<br>##)<br>Change | CCX168<br>Standar<br>(N= | d of Care | All<br>(N= | CCX168<br>##)<br>Change |
|---|---|---|---|---|---|---|---|---|
| Parameter 1 (U | Jnit) | | | | | | | |
| Baseline | | | | | | | | |
| N' | ** | | ** | | ** | | ** | |
| Mean | **-* | | **-* | | **-* | | **** | |
| SD | **.** | | **.** | | **.** | | **.** | |
| SEM | **.** | | **.** | | **.** | | **.** | |
| Minimum | ** . | | ** . | | ** . | | ** . | |
| Median | **.* | | **.* | | **.* | | **.* | |
| Maximum | ** | | ** | | ** | | ** | |
| Day 2 | | | | | | | | |
| N' | 44 | ## | ** | ** | ** | ## | 44 | 0.6 |
| Mean | 44.4 | 80.8 | **.* | 80.8 | **.* | 80.8 | 44.4 | 48.4 |
| SD | **.** | ##.## | **.** | ##.## | **.** | ##.## | 11.11 | 99.99 |
| SEM | **.** | **.** | **.** | **.** | **.** | **.** | **.** | **.** |
| Minimum | ** | ## | ** | ## | ** | ## | 6.6 | 0.6 |
| Median | **.* | ##.# | **.* | **.* | **.* | **.* | **.* | 99.9 |
| Maximum | ** | ** | ** | ** | ** | ** | ** | ** |

The vital sign parameters to be summarized include:

Systolic blood pressure, Diastolic blood pressure, Heart rate, Oral temperature, Weight, BMI.

The visits to be summarized include:

Day 2, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, End of Treatment, Day 99, Day 113, Day 141, Day 169, End of Follow-up Period for systolic blood pressure, diastolic blood pressure, heart rate, and oral temperature, and Day 15, Day 29, Day 57, Day 85, End of Treatment, Day 113, Day 169, and End of Follow-up Period for Weight and BMI.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

<sup>-</sup> Baseline is defined as the last pre-dose value.

<sup>-</sup> N'=number of subjects with data at baseline and the specified visit.

<sup>-</sup> The End of Treatment value is the last measurement through Day 85.

<sup>-</sup> The End of Follow-up Period is the last measurement after Day 85 through Day 169.

#### Table 14.3.5.2 Summary of Physical Examination and Body System Reviews by Visit Safety Population

| Day | | | | bo +<br>of Care | | | 10 mg +<br>of Care | | | 0 mg +<br>of Care | | 1 CCX | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Body System | Result | N' | n | (%) | N' | n | | N' | n | (%) | N' | n | (%) |
| Day 1 | | | | | | | | | | | | | |
| General Appearance | Normal/same as previous PE<br>Abnormal, new since previous PE | | | (###.#)<br>(###.#) | | ** | (###.#)<br>(###.#) | ** | ** | (###.#)<br>(###.#) | | ** | (###.# |
| HEENT | Normal/same as previous PE<br>Abnormal, new since previous PE | | ** | (###.#)<br>(###.#) | ** | ** | (###.#)<br>(###.#) | ** | ** | (###.#)<br>(###.#) | | ** | (###.<br>(###. |

The body systems to be summarized include:

General Appearance/Mental Status, HEENT, Dermatologic, Cardiovascular, Respiratory, Gastrointestinal, Musculoskelatal, and Dermatologic.

The visits to be summarized include:

Day 1, Day 2, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113, Day 141, and Day 169.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

<sup>-</sup> N'=number of subjects with body system reviewed at the specified visit.


## Table 14.3.5.3 Listing of ECG Abnormalities Safety Population

| Treatment<br>Subject Age/Sex/Race | Date/Day | Abnormality | Clinically<br>Significant? |
|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX DDMMMYYYY/XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY

NOTE: This table will be sorted by treatment group and subject within treatment group.

| 8 Listing Shells | |
|---|---|
| Listing D1 | 108 |
| Subject Treatment Information, Demographics, and Baseline Characteristics | |
| All Randomized Subjects | |
| Listing D2 | 109 |
| Study Medication Information | |
| All Randomized Subjects | |
| Listing D3.1 | 110 |
| Cyclophosphamide IV Dosing | |
| All Randomized Subjects | |
| Listing D3.2 | 111 |
| Rituximab Dosing (Step 3) | |
| All Randomized Subjects | |
| Listing D4 | 113 |
| Concomitant Medications | |
| All Randomized Subjects | |
| Listing D5 | 114 |
| Adverse Events | |
| All Randomized Subjects | |
| Listing D6 | 115 |
| Central Laboratory Data - Chemistry | |
| All Randomized Subjects | |
| Listing D7 | 116 |
| Central Laboratory Data - Hematology | |
| All Randomized Subjects | |
| Listing D8 | 116 |
| Central Laboratory Data - Urinalysis | |
| All Randomized Subjects | |
| Listing D9 | 116 |
| Central Laboratory Data – Urine Chemistry | |
| All Randomized Subjects | |
| Listing D10.1 | 116 |
| Local Laboratory Data - Serum Chemistry, Hematology, and Coagulation | |
| All Randomized Subjects | |
| Listing D10.2 | 116 |
| Local Laboratory Data – Virology, Immunology, and Chest X-ray Results | |
| All Randomized Subjects | |
| Listing D11 | 117 |
| Local Laboratory Data - Urinalysis | |
| All Randomized Subjects | |
| Listing D12 | 118 |
| Birmingham Vasculitis Activity Score (BVAS) | |
| All Randomized Subjects | |

| Listing D13 | 119 |
|-----------------------------------------------------------------------|-----|
| Vasculitis Damage Index | |
| All Randomized Subjects | |
| Listing D14 | 120 |
| ANCA Results | |
| All Randomized Subjects | |
| Listing D15 | 121 |
| Serum hsCRP Results (mg/L) | |
| All Randomized Subjects | |
| Listing D16 | 122 |
| Serum Urinary MCP-1:Creatinine Ratio Results (pg/mg Creatinine) | |
| All Randomized Subjects | |
| Listing D17 | 123 |
| Estimated Glomerular Filtration Rate (MDRD) Results (mL/min/1.73 m^2) | |
| All Randomized Subjects | |
| Listing D18 | 124 |
| ACR Results (mg/g) | |
| All Randomized Subjects | |
| Listing D19 | 125 |
| Vital Signs, Weight, and BMI | |
| All Randomized Subjects | |
| Listing D20 | 126 |
| Physical Exam and Body System Reviews | |
| All Randomized Subjects | |
| Listing D21 | 127 |
| SF-36v2 Health Survey | |
| All Randomized Subjects | |
| Listing D22 | 129 |
| EQ-5D-5L Questionnaire and VAS | |
| All Randomized Subjects | |


#### Listing D1 Subject Treatment Information, Demographics, and Baseline Characteristics All Randomized Subjects

SUBJECT: ###-###

#### TREATMENT INFORMATION

Treatment: CCX168

Date of First Dose: DDMMMYYYY Date of Last Dose (Day): Ongoing

Date of Completion/Early Termination (Day): Ongoing

Did the Subject Complete the Study?: No

#### BASELINE INFORMATION

Protocol version: Amendment #

Body weight (kg): ##.# BMI (kg/m^2): ##.#

Smoking status: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX AAV Status: (Specify as newly diagnosed or relapsed.)

Date of AAV Diagnosis: DDMMMYYYY Duration of AAV disease: ##.#

Type of AAV: (Specify as Granulomatosis with polyangiitis (Wegener's), Microscopic polyangiitis, or Renal limited vasculitis)

IIF Test for P-ANCA: (Specify as positive or negative.) IIF Test for C-ANCA: (Specify as positive or negative.)

ELISA Test for Anti-proteinase-3: (Specify as positive or negative.) ELISA Test for Anti-myeloperoxidase: (Specify as positive or negative.)

Baseline Birmingham Vasculitis Activity Score (BVAS): ##

Baseline Vasculitis Damage Index Score (VDI): ##

Was renal biopsy done to confirm diagnosis of renal vasculitis? XXX [If yes, describe abnormalities.]

Baseline Estimated Glomerular Filtration Rate (MDRD) Results (mL/min/1.73 m^2): ##.#

Baseline ACR (mg/g): ##.#

Baseline Urine Red Blood Cell Count (/hpf): ##

Baseline MCP-1:Creatinine Ratio(pg/mg Creatinine): ##

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM
#### Listing D2 Study Medication Information All Randomized Subjects

| Treatment<br>Subject | Visit | Date | | pensed Capsules Returned | | ednisone<br>ed Tablets Returned |
|---|---|---|---|---|---|---|
| (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | OXXXXXXXXXXX | XXXXXX | | | | |
| ***-*** | Day 1<br>Day 8<br>Day 15 | DDMMMYYYY<br>DDMMMYYYYY<br>DDMMMYYYYY | ** | ** | ** | ** |
| | Overall | of Dosing (days):<br>Percent Compliance<br>X168 or Prednisone | :: | ***.* | *** | +.+ |
| 0000000000000 | 0000000000 | XXXXXXX | | | | |
| ***-*** | Day 1<br>Day 8<br>Day 15 | DDMMMYYYY<br>DDMMMYYYYY<br>DDMMMYYYYY | ** | ** | ** | ** |
| | Overall | of Dosing (days):<br>Percent Compliance<br>X168 or Prednisone | 1: | *** | *** | 1.1 |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

Note to programmer: For the calculation of prednisone dose, most subjects used bottles containing 20 mg prednisone for the first week and then bottles containing 5 mg prednisone after week 1 (refer to protocol section 11.6 for details).

## Listing D3.1 Cyclophosphamide IV Dosing All Randomized Subjects

| Treatment | | | Was Cyclophosphamide<br>Administered | Dose Aministered | Total Dose Aministered |
|---|---|---|---|---|---|
| | *** | D | | | |
| Subject | Visit | Date | At This Visit? | (mg/kg) | (mg) |
| OXXXXXXXXXXX | xxxxxxxxx | xxxxx | | | |
| ***-*** | Day 1 | DDMMMYYYY | XXX | *** | |
| | Day 15 | DDMMMYYYY | XXX | *** | *** |
| | Day 29 | DDMMMYYYY | XXX | *** | *** |
| | Day 57 | DDMMMYYYY | XXX | *** | 111 |
| | Day 85 | DDMMMYYYYY | XXX | *** | *** |
| | - | | | | |
| | Total Da | ys of Dosing D | buring 84-Day Treatment Peri | od: | *** |
| | | | Treatment Period: | | *** |
| | Day 113 | DDMMMYYYY | XXX | *** | *** |
| | Day 141 | DDMMMYYYYY | XXX | *** | *** |
| | Day 169 | DDMMMYYYY | XXX | *** | *** |
| | 227 203 | | | 200 | |
| | Total Da | vs of Dosing D | ouring 168-Day Treatment Per | iod: | *** |
| | | | y Treatment Period: | | *** |

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYYY HH:MM

### Listing D3.2 Rituximab Dosing All Randomized Subjects

| Treatment<br>Subject | Visit | Date | Was Rituximab<br>Administered<br>At This Visit? | Start Date/Time | Stop Date/Time | Total Dose<br>Aministered<br>(mg) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|
| OXXXXXXXXXX | | | | P. P | P. 100 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | waaaaaaaaaaaa |
| ***-*** | Day 1 | DDMMMYYYYY | XXX | DDMMMYYYY/HH:MM | DDMMYYYY/HH:MM | *** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | XXX<br>XXX | DDMMYYYY/HH:MM<br>DDMMMYYYY/HH:MM<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM<br>DDMMMYYYY/HH:MM<br>DDMMMYYYY/HH:MM | *** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM


Listing D3.3 Oral Azathioprine Dosing All Randomized Subjects

VISIT: Day 1 DATE: MMDDYYYY -----

Azathioprine initiated at this visit?: XXX Start date/Stop date: DDMMMYYYY/DDMMMYYYY

Initial dose administered (mg): ###

Was target dose of 2 mg/kg/day reached: XXX

If yes, date: DDMMMYYYY Total daily dose: ###

If no, maximum daily dose administered: XXX

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM


Listing D4 Concomitant Medications All Randomized Subjects

RT: Reported Term

ATC: Anatomic Therapeutic Class Start Date (Day) / Treatment

PT: Preferred Term End Date (Day) Dose/Unit Frequency Subject Route

\*\*\*-\*\*\* DDMMMYYYY (###)/ 

DDMMMYYYY (###)

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM


## Listing D5 Adverse Events All Randomized Subjects

| Treatment<br>Subject | TEAE? | RT: Reported Term<br>OC: Primary System Organ Class<br>PT: Preferred Term | Start Date (Day)<br>End Date (Day) | | Related-<br>ness[1] | | | Improve/<br>Disappear[5] | Reappear/ |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (###)/<br>DDMMMYYYY (###) | XXXXXXXXX | */*/* | • | */* | хх | хх |

- An adverse event is considered treatment-emergent if the start date of the event is on or after administration of the first dose of study medication. 'Day' is the number of days from the date of randomization.
- [1] Relatedness: (Study Medication/Corticosteroid/Cyclophosphamide) 0=Probably Not Related, 1=Possibly Related
- [2] Actions Taken: 1-None, 2-Study medication discontinued, 3-Study medication interrupted
- [3] Outcome: 1=Resolved, 2=Resolved with sequelae, 3=Ongoing, 4=Death, 5=Unknown
- [4] Serious Outcome: 1=Results in death, 2=Life threatening, 3=Inpatient hospitalization or prolongation of existing hospitalization, 4=Persistent or significant disability/incapacity, 5=Congenital abnormality or birth defect, 6=Important medical event
- [5] Did the event improve or disappear after stopping study medication (dechallenge)?
- [6] Did the event reappear or worsen after restarting study medication (rechallenge)?

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM


### Listing D6 Central Laboratory Data - Chemistry All Randomized Subjects

Abnormal Treatment Normal Subject Parameter (Unit) Range Visit Value Flag

\*\*\*\*\*\*\*\*\*\* NOTABLE HIGH

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY The following listings will have the same layout as Listing D6:

Listing D7 Central Laboratory Data - Hematology All Randomized Subjects

Listing D8 Central Laboratory Data - Urinalysis All Randomized Subjects

Listing D9
Central Laboratory Data - Urine Chemistry
All Randomized Subjects

Listing D10.1

Local Laboratory Data - Serum Chemistry, Hematology, and Coagulation
All Randomized Subjects

Listing D10.2

Local Laboratory Data - Virology, Immunology, and Chest X-ray Results
All Randomized Subjects

Note to programmer: Verify the contents of this table with data management.


## Listing D11 Local Laboratory Data - Urinalysis All Randomized Subjects

| Subject | Treatment | Sample<br>Collected? | RBC<br>Count<br>(/hpf) | RBC<br>Casts | Any<br>Clots<br>Present? | Was Transfusion Required/<br>Any Urinary Tract Obstruction? |
|---|---|---|---|---|---|---|
| ****-*** | XXXXXXXXXXXXXXXXXXXXXXX | xxx | *** | xxxxxxx | xxx | xxx |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMYYYYY

## Listing D12 Birmingham Vasculitis Activity Score (BVAS) All Randomized Subjects

| Subject | Treatment | Visit | Date | Was<br>BVAS<br>Assessed? | Category | Baseline<br>Score | Visit<br>Score | Change<br>from<br>Baseline | <pre>&amp; Change from Baseline</pre> |
|---|---|---|---|---|---|---|---|---|---|
| 111-111 | XXXXXXXXXX | Screening | DDMMMYYYY | Yes | General Cutaneous Mucous membrane/eyes Ear, nose, throat Chest Cardiovascular Abdominal Renal Nervous system Other BVAS Total | ** | ** | ** | 11.1 |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

## Listing D13 Vasculitis Damage Index All Randomized Subjects

| Subject | Treatment | Visit | Date | Was<br>VDI<br>Assessed? | Category | Baseline<br>Score | Visit<br>Score | Change<br>from<br>Baseline | <pre>\$ Change from Baseline</pre> |
|---|---|---|---|---|---|---|---|---|---|
| 111-111 | XXXXXXXXX | Screening | DDMMYYYY | Yes | Musculoskelatal Skin/Mucous membra Ocular ENT Pulmonary Cardiovascular PVD Gastrointestinal Renal Neuropsychiatric Other Overall VDI Score | ## | ** | " | 11.1 |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

## Listing D14 ANCA Results All Randomized Subjects

| Subject | Treatment | Visit | Date | Parameter | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline | % Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| ***-** | xxxxxxxx | Screening | DDMMMYYYY | Anti-PR3 (IU/mL)<br>Anti-MPO (IU/mL) | ** | ** | ** | 11.1 |

- Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

### Listing D15 Serum hsCRP Results (mg/L) All Randomized Subjects

| Subject | Treatment | Visit | Date | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline | % Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|
| ***-** | XXXXXXXXX | Screening | DDMMYYYY | ** | ** | ** | **-* |

<sup>-</sup> Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYYY HH:MM


### Listing D16 Serum Urinary MCP-1:Creatinine Ratio Results (pg/mg Creatinine) All Randomized Subjects

| Subject | Treatment | Visit | Date | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline | % Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|
| ***-** | XXXXXXXXXX | Screening | DDMMMYYYY | ** | ** | ** | **-* |

<sup>-</sup> Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM


# Listing D17 Estimated Glomerular Filtration Rate (MDRD) Results (mL/min/1.73 m^2) All Randomized Subjects

| Subject | Treatment | Visit | Date | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline | <pre>% Change from Baseline</pre> |
|---|---|---|---|---|---|---|---|
| ***-*** | xxxxxxxx | Screening | DDMMMYYYY | ** | ** | ** | **-* |

- Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM

### Listing D18 ACR Results (mg/g) All Randomized Subjects

| Subject | Treatment | Visit | Date | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline | % Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|
| ***-** | XXXXXXXXX | Screening | DDMMYYYY | ** | ** | ** | **-* |

<sup>-</sup> Baseline is defined as the last pre-dose value.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYYY HH:MM


## Listing D19 Vital Signs, Weight, and BMI All Randomized Subjects

| Subject | Treatment | Visit | Date | Parameter | Baseline<br>Result | Visit<br>Result | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|
| 111-111 | XXXXXXXXX | Screening | DDMMMYYYY | Systolic Blood Pressure (mmHg) Diastolic Blood Pressure (mmHg) Heart Rate (bpm) Oral Temperature (F) Height (cm) Weight (kg) Body Mass Index (kg/m^2) | ** | ** | ** |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMYYYY HH:MM

## Listing D20 Physical Exam and Body System Reviews All Randomized Subjects

| Subject | Treatment | Visit | Date | Body System | Result | Abnormal Finding(s) |
|---|---|---|---|---|---|---|
| ***-*** | 2000000000 | Screening | DDMMYYYY | General Apperance/Mental Status<br>HEENT<br>Dermatologic<br>Cardiovascular<br>Respiratory<br>Gastrointestinal<br>Musculoskeletal<br>Neurologic | Not done<br>Normal<br>Normal<br>Normal<br>Normal<br>Normal<br>Abnormal | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Database last modified: DDMMYYYYY HH:MM


Listing D21 SF-36v2 Health Survey All Randomized Subjects

XXXXXXXXXXXXXXXXXXXXXXX

XXXXXXXXXXXXXXXXXXXXXXXX

VISIT: Day 1 DATE: MMDDYYYY

In general, would you say your health is:

Compared to one year ago, how would you rate your health in general now:

How much does your health now limit you in the following activities:

Vigorous activities:

Moderate activites:

Lifting of carrying grocieries:

Climbing several flights of stairs:

Climbing one flight of stairs:

Bending, kneeling, or stooping:

Walking more than a mile:

Walking several hundred yards:

Walking one hundred yards:

Bathing or dressing yourself:

During the past 4 weeks, how much of the time have you had problems with the following as a result of your physcial health:

Cut down on the amount of time you spent on work or other activities:

Accomplished less than you would like:

Were limited in the kind of work or other activities:

Had difficulty performing the work or other activities:

During the past 4 weeks, how much of the time have you had problems with the following as a result of your emotional health:

Cut down on the amount of time you spent on work or other activities:

Accomplished less than you would like:

Did work or other activities less carefully than usual:

During the past 4 weeks, to what extent has physical or emotional health interfered with social activites:

How much bodily pain have you had in the last 4 weeks:

During the past 4 weeks, how much did pain interfere with your normal work:

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM


Listing D21 SF-36v2 Health Survey All Randomized Subjects

VISIT: Day 1 DATE: MMDDYYYY During the past 4 weeks: Did you feel full of life: Have you been very nervous: Have you felt so down in the dumps that nothing could cheer you up: Have you felt calm and peaceful: Did you have a lot of energy: Have you felt downhearted and low: Did you feel worn out: Have you been happy: Did you feel tired: During the past 4 weeks, how much of the time has your physical or emotional problems interfered with your social activities: How TRUE or FALSE is each of the following statements for you: I seem to get ill more easily than other people I am as healthy as anybody I know: I expect my health to get worse: My health is excellent: Summary Scores: Role-Physical: Role-Emotional: Social Functioning: Bodily Pain: Mental Health: General Health Perceptions: Change in Health: Physcial Component Summary: Mental Health Summary:

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM

### Listing D22 EQ-5D-5L Questionnaire and VAS All Randomized Subjects

| Subject Treatment Visit Date Question Result ###-### XXXXXXXXXXX Day 1 DDMMYYYY Mobility Self-care Usual activities Pain/Discomfort Anxiety Depression Health Scale Score VAS | | | | | | |
|---|---|---|---|---|---|---|
| Self-care Usual activities Pain/Discomfort Anxiety Depression Health Scale Score | Subject | Treatment | Visit | Date | Question | Result |
| | ***-*** | XXXXXXXXXXX | Day 1 | DDMMYYYY | Self-care Usual activities Pain/Discomfort Anxiety Depression Health Scale Score | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Database last modified: DDMMMYYYY HH:MM


Listing D23 Renal Biopsy Histology All Randomized Subjects

DATE OF BIOPSY: MMDDYYYY

Observations based on light miscoscopy:

Arteritis in biopsy? XXXXXXXXXXXXXXXXXXXXXXXX

Database last modified: DDMMYYYY HH:MM Program Name: XXXXXXXX.sas Run Date: DDMMMYYYYY HH:MM

Note to programmer: Only display data for biopsies performed.